

Title: A Phase 2, Open-Label, Multicenter Study of Ixazomib Plus Lenalidomide and Dexamethasone in Adult Japanese Patients With Relapsed and/or Refractory Multiple Myeloma

NCT Number: NCT02917941

Statistical analysis plan Approve Date: 19-SEP-2018

Certain information within this statistical analysis plan has been redacted (ie, specific content is masked irreversibly from view with a black/blue bar) to protect either personally identifiable information or company confidential information.

This may include, but is not limited to, redaction of the following:

- Named persons or organizations associated with the study.
- Patient identifiers within the text, tables, or figures or in by-patient data listings.
- Proprietary information, such as scales or coding systems, which are considered confidential information under prior agreements with license holder.
- Other information as needed to protect confidentiality of Takeda or partners, personal information, or to otherwise protect the integrity of the clinical study.

If needed, certain appendices that contain a large volume of personally identifiable information or company confidential information may be removed in their entirety if it is considered that they do not add substantially to the interpretation of the data (eg, appendix of investigator's curriculum vitae).



### STATISTICAL ANALYSIS PLAN

**STUDY NUMBER: C16028** 

3. Policable Terms of Use A Phase 2, Open-Label, Multicenter Study of Ixazomib Plus Lenalidomide and Dexamethasone in Adult Japanese Patients With Relapsed and/or Refractory Multiple Myeloma

### PHASE 2

Version: 2 Date: 19 September 2018

Prepared by:

PPD

PPD

Based on:

Protocol Version: Amendment 1 Protocol Date: 25 November 2016

### CONFIDENTIAL PROPERTY OF TAKEDA

This document is a confidential communication of Takeda. Acceptance of this document constitutes the agreement by the recipient that no information contained herein will be published or disclosed without written authorization from Takeda.



# 2.0 TABLE OF CONTENTS

| 1.0 | | | E PAGE | |
|---|---|---|---|---|
| | 1.1 | | pproval Signatures | |
| 2.0 | | TABL | E OF CONTENTSOF ABBREVIATIONS | <sub>.</sub> 3 |
| 3.0 | | LIST | OF ABBREVIATIONS | ك5 |
| 4.0 | | OBJE | CTIVES | 7 |
| | 4.1 | Pr | CTIVES imary Objectives condary Objectives dditional Objectives | 7 |
| | 4.2 | Se | condary Objectives | 7 |
| | 4.3 | Ac | lditional Objectives | 7 |
| | 4.4 | St | udy Design | 7 |
| 5.0 | | ANAI | LYSIS ENDPOINTS | 9 |
| 6.0 | | DETE | RMINATION OF SAMPLE SIZE | 9 |
| 7.0 | | METH | udy Design LYSIS ENDPOINTS RMINATION OF SAMPLE SIZE | 10 |
| | 7.1 | Ge | Study Definitions Definition of Study Visit Windows | 10 |
| | | 7.1.1 | Study Definitions | 10 |
| | | 7.1.2 | Definition of Study Visit Windows | 11 |
| | | 7.1.3 | Significance Level and Confidence Coefficient | 11 |
| | 7.2 | Ar | Significance Level and Confidence Coefficient | 11 |
| | 7.3 | Di | sposition of Subjects | 12 |
| | | 7.3.1 | Study Information | 12 |
| | | 7.3.2 | Number of Subjects Who Entered the Treatment Period by Site | 12 |
| | | 7.3.3 | Disposition of Subjects | 12 |
| | | 7.3.4 | Protocol Deviations and Analysis Sets | 13 |
| | 7.4 | De | emographic and Other Baseline Characteristics | 14 |
| | 7.5 | Me | edical History and Concurrent Medical Conditions | 22 |
| | 7.6 | Me | edication History and Concomitant Medications | 23 |
| | 7.7 | St | udy Drug Exposure and Compliance | 23 |
| | 7.8 | Ef | ficacy Analysis | 26 |
| | ( | 7.8.1<br>7.8.2 | Primary Efficacy Endpoint(s) | 26 |
| 1 | St. | 7.8.2 | Secondary Efficacy Endpoint(s) | 27 |
| | | 7.8.3 | Additional Efficacy Endpoint(s) | 30 |
| )` | | 7.8.4 | Statistical/Analytical Issues | 32 |
| | 7.9 | Ph | armacokinetic/Pharmacodynamic Analysis | 35 |
| | | 7.9.1 | Pharmacokinetic Analysis | 35 |
| | | 7.9.2 | Pharmacodynamic Analysis | 35 |
| | 7.1 | 0 Ot | her Outcomes | 35 |
| | 7.1 | 1 Sa | fety Analysis | 36 |
| | | 7.11.1 | Adverse Events | 36 |

### 3.0 LIST OF ABBREVIATIONS

5-HT3

ADL

ΑE

ALT **ANC** AST

anization

graphy

alon

deoxyribonucleic acid
duration of response
Eastern Cooperative Oncology Group
electronic case report form
and of Treatment (visit)
ill analysis set
nale patients of childbesited States Food
rescent in Fight **BUN** CBC CI  $CO_2$ CR

**CRO** 

CT **CYP** 

Del

**DNA** DOR

**ECOG** 

eCRF **EOT FAS** 

**FCBP FDA** 

**FISH** 

free light chain **FLC** Good Clinical Practice **GCP** 

granulocyte colony stimulating factor G-CSF

**GVHD** graft-versus-host disease **HBcAb** hepatitis B core antibody

**HBV** hepatitis B virus ъв ICH IMir **HCV** hepatitis C virus

human immunodeficiency virus

Investigator's Brochure

International Conference on Harmonisation

immunomodulatory drugs

**IMWG** International Myeloma Working Group

IRB institutional review board **ISS** international staging system

IUD intrauterine device

IV intravenous; intravenously lenalidomide and dexamethasone LenDex

LDH lactate dehydrogenase

MedDRA Medical Dictionary for Regulatory Activities

### C16028 Statistical Analysis Plan Version 2

**MHRA** Medicines and Healthcare products Regulatory Agency

MM multiple myeloma

MRI magnetic resonance imaging

NCI CTCAE National Cancer Institute Common Terminology Criteria for Adverse Events

**NDMM** newly diagnosed multiple myeloma

ORR overall response rate OS overall survival

PD progressive disease (disease progression)

PET positron emission tomography **PFS** progression-free survival

**PMDA** Pharmaceuticals and Medical Devices Agency **PML** progressive multifocal leukoencephalopathy

applicable Terms of Use my progressive municipal reukoencephalopathy polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin **POEMS** 

changes

PR partial response

**PRES** posterior reversible encephalopathy syndrome.

PTE pretreatment event RNA ribonucleic acid

relapsed and/or refractory multiple myeloma **RRMM** 

SAE serious adverse event SAP statistical analysis plan sCR stringent complete response

stable disease SD

**SPEP** serum protein electrophoresis

**SUSAR** suspected unexpected serious adverse reaction

**TEAE** treatment-emergent adverse event TEN toxic epidermal necrolysis

time to first occurrence of maximum (peak) concentration  $T_{\text{max}}$ 

**TSH** thyroid stimulating hormone

TTP time to progression

ULN upper limit of the normal range urine protein electrophoresis very good partial response

white blood cell

World Health Organization

### 4.0 **OBJECTIVES**

10 determine VGPR or better (VGPR + CR) rate in response-evaluable analysis set\*

\*Defined as patients who received at least one dose of ixazomib and had measurable disease at baseline, and at least one post baseline response assessment.

4.2 Secondary Objectives

• To determine progression-free survival (PFS)

• To determine overall response rate (ORR) (partial response [PR] or better)

• To determine duration of response (DOR)

• To determine time to progression (TTD)

- To determine safety
- To determine overall survival (OS)

### 4.3 **Additional Objectives**

Not applicable

### 4.4 **Study Design**

only and subject to the ic This is a phase 2, open-label, single arm, multicenter study to evaluate the efficacy and safety of ixazomib plus lenalidomide and dexamethasone in Japanese patients with relapsed and/or refractory multiple myeloma (MM). The patient population will consist of adult men and women who have a confirmed diagnosis of MM, who have received 1 to 3 prior lines of therapy, and who meet other outlined eligibility criteria (see Section 7.0). Approximately 30 patients will be enrolled in the study.

General eligibility criteria may be assessed prior to the formal Screening period if it is part of standard clinical practice. However, per the Schedule of Events, formal screening will occur during the Screening period, which may last for up to 28 days prior to enrollment. A Takeda clinician will confirm patient eligibility prior to enrollment. Determination of disease progression as an entry criterion may be based on patient data obtained during or following the patient's most recent prior antineoplastic therapy.

Patients will receive study drug (ixazomib 4.0 mg) on Days 1, 8, and 15 plus lenalidomide (25 mg) on Days 1 through 21 and dexamethasone (40 mg) on Days 1, 8, 15, and 22 of a 28day cycle. Patients may continue to receive treatment until progressive disease (PD) or unacceptable toxicity, whichever comes first. Dose modifications may be made based on toxicities. Patients with a low creatinine clearance < 60 mL/min will receive a reduced lenalidomide dose of 10 mg. The lenalidomide dose may be escalated to 15 mg after 2 cycles if the patient is not responding to treatment and is tolerating the treatment. If renal function normalizes (ie, creatinine clearance ≥ 60 mL/min) and the patient continues to tolerate this treatment, lenalidomide may then be escalated to 25 mg.

Patients will be seen at regular treatment cycle intervals while they are participating in the study: four times a treatment cycle for the first 2 cycles, twice a treatment cycle for the 3rd

150 NSE

cycle, and then once a treatment cycle for the remainder of their participation in the active treatment and, if applicable, the PFS (every 4 weeks) and OS (every 12 weeks) follow-up phases of the study.

Response will be assessed by investigator according to the IMWG criteria for all patients every 4 weeks until PD. Central laboratory data will be used for serum M-protein, urine M-protein and serum free light chain. All patients will be followed for survival after progression. Patients will be contacted every 12 weeks until death or termination of the study by the sponsor.

Patients will attend an End of Treatment (EOT) visit approximately 30 days after receiving their last dose of study treatment (ixazomib, lenalidomide or dexamethasone) and will continue to be followed for other follow-up assessments specified in the Schedule of Events. Patients discontinuing study treatment prior to PD will continue to be assessed for PD during the PFS follow-up portion of the study.

Analysis is planned to be performed twice during the study. The primary analysis is planned to be performed using the data obtained at approximately 12 months from the enrollment of the last patient. The final analysis is planned to be performed after the final database lock en ational at a seed a for non-commercial use only all a property of Takeda. For non-commercial use only a seed a for non-commercial use only a seed a se using the data obtained at approximately 24 months from the enrollment of the last patient. The timing of analysis may be changed or additional analysis may be added upon request of

### 5.0 ANALYSIS ENDPOINTS

### Primary Efficacy Endpoint

VGPR or better rate in response-evaluable analysis set

### Secondary Efficacy Endpoints

- PFS, defined as the time from the date of first study drug administration to the date of first documentation of PD or death from any cause, whichever occurs first
- ORR
- DOR, defined as the time from the date of first documentation of response to the date of first documentation of PD
- TTP, defined as the time from the date of first study drug administration to the date of first documentation of PD
- Safety including treatment-emergent adverse events (TEAEs), laboratory parameters, and vital signs
- OS, defined as the time from the date of first study drug administration to the date of death

# 6.0 DETERMINATION OF SAMPLE SIZE

Assuming the expected VGPR or better rate is 48.1% and the threshold rate is 39.0% based on the results of Study C16010, a sample size of 27 would be necessary to provide a point estimate of VGPR or better rate higher than the threshold rate with 80% probability. Assuming a drop-out ratio of 10%, the target number of patients has been set to 30. The expected response rate and the threshold assumptions are based on VGPR or better rate in ixazomib + LenDex arm and placebo + LenDex arm in Study C16010 (intent-to-treat population, primary analysis).

### 7.0 METHODS OF ANALYSIS AND PRESENTATION

# 7.1 General Principles

### 7.1.1 Study Definitions

The following definitions and calculation formulas will be used.

- Descriptive statistics: Number of subjects, mean, standard deviation, maximum, minimum, and quartiles
- Frequency distributions: Number of subjects and percentage (of nonmissing) percategory
- Baseline body surface area (m<sup>2</sup>): square root of (baseline height \* baseline weight / 3600)
- Time since initial diagnosis to first dose at study entry (months): (first dose date date of initial diagnosis + 1) / (365.25 / 12)
- Relapsed patients: Patients who relapsed from at least 1 previous treatment but were not refractory to any previous treatment. Patients who progress after 60 days from the last dose of a given therapy will be considered relapsed.
- Refractory patients: Patients who were refractory to at least 1 previous treatment but were not relapsed to any previous treatment. Refractory disease is defined as disease progression on treatment or progression within 60 days after the last dose of a given therapy.
- Refractory and relapsed patients: Patients who were relapsed from at least 1 previous treatment and additionally were refractory to at least 1 previous treatment.
- Primary refractory patients: Patients who are refractory to all lines of previous therapy (i.e., best response to prior therapy is SD or disease progression on all lines of therapy).
- Time since last transplant to first dose at study entry (months): (first dose date start date of prior transplant) / (30.4375)
- Relative dose intensity: 100 \* (total amount of dose taken) / (total prescribed dose of treated cycles), where total prescribed dose equals [dose prescribed at enrollment \* number of prescribed doses per cycle \* the number of treated cycles]
- Extent of Exposure (cycles) is based on the number of treated cycles.
- Extent of Exposure (days): date of last dose date of first dose + 1
- Percent drug compliance (%): (study drug taken in mg) / (study drug expected to be taken in mg) \*100%
- Treatment-emergent adverse event (TEAE): Any adverse event that occurs after administration of the first dose of any study drug through 30 days after the last dose of any study drug
- If corrected calcium is not reported directly, it can be calculated using the following formula:
  - ➤ Corrected Calcium (mmol/L): serum calcium (mmol/L) + 0.0200 \* (40 serum albumin (g/L))

### **Definition of Study Visit Windows**

Ablicable Leiths of Use Unless otherwise specified, the baseline value is defined as the value collected at the time closest to, but before, the start of study drug administration.

All data will be categorized on the basis of the scheduled visit at which they are collected.

### 7.1.3 Significance Level and Confidence Coefficient

Confidence coefficient: 95% (two-sided)

### 7.2 **Analysis Sets**

In this study, the following three analysis sets are defined.

- FAS: All subjects who received at least one dose of the study drug during the treatment period. Subjects will be excluded from FAS if the following criterion is met:
  - No study drug received
- Response-evaluable analysis set: All FAS subjects with measurable disease at baseline, and at least one post baseline response assessment. Measurable disease is defined by at least 1 of the following 3 measurements based on central laboratory data: serum Mprotein  $\ge 1$  g/dL ( $\ge 10$  g/L), urine M-protein  $\ge 200$  mg/24 hours, and serum free light chain assay where involved free light chain level≥10 mg/dL (≥ 100 mg/L), provided that the serum free light chain ratio is abnormal.

Subjects will be excluded from the response-evaluable analysis set if any of the following criteria are met:

- No measurable disease at baseline
- No post-baseline assessment
- No study drug received
- Safety analysis set: All subjects who received at least one dose of the study drug during the treatment period. Subjects will be excluded from the safety analysis set if the following criterion is met:
- Property of Lakeda No study drug received

# 7.3 Disposition of Subjects

### 7.3.1 Study Information

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis

Variable(s): Date First Subject Signed Informed Consent Form

Date of Last Subject's Last Visit/Contact

MedDRA Version
WHO Drug Version

SAS Version Used for Creating the Datasets

Analytical

Method(s): (1) Study Information

Study information shown in the analysis variables section will be provided.

### 7.3.2 Number of Subjects Who Entered the Treatment Period by Site

Analysis Set: All Subjects Who Entered the Treatment Period

Analysis

Variable(s): Status of Entrance into the Treatment [Entered]

Period

Stratum: Site [Site numbers will be used as

categories]

Analytical

Method(s): (1) Number of Subjects Who Entered the Treatment Period by Site

Frequency distribution will be provided for each stratum.

### 7.3.3 Disposition of Subjects

Analysis Set: All Subjects Who Entered the Treatment Period

Analysis

Variable(s): Study Drug Completion Status [Ongoing on Treatment, Prematurely

Discontinued Study Drug]

Reason for Discontinuation of [Adverse Event, Lost to Follow-up,

Study Drug Progressive Disease, Protocol

Violation, Study Terminated by Sponsor, Withdrawal by Subject,

Other]

Subjects that have Participated in OS

Follow-up

Subjects that have Participated in [Yes, No]

PFS Follow-up

Completion Status of the Follow-up [Completed Follow-up Period,

Period Prematurely Discontinued Follow-up

Period]

Reason for Discontinuation of the [Lost to Follow-up, Study Terminated

Follow-up Period by Sponsor, Withdrawal by Subject,

Other

Analytical

Method(s): (1) Disposition of Subjects

Frequency distributions will be provided.

### 7.3.4 Protocol Deviations and Analysis Sets

### 7.3.4.1 Protocol Deviations

Analysis Set: All Subjects Who Entered the Treatment Period

**Analysis** 

Variable(s): Significant Protocol [Entry Criteria, Concomitant Medication,

Deviation Procedure Not Performed Per Protocol, Study

Medication, Withdrawal Criteria, Good Clinical

Practice]

Analytical

Method(s): (1) Protocol Deviations

Frequency distribution will be provided for each deviation category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be classified into the

same category will be counted only once.

7.3.4.2 Analysis Sets

Analysis Set: All Subjects Who Entered the Treatment Period

Analysis

Variable(s): Handling of Subjects [Categories are based on the

specifications in Section 7.2

Analytical

Method(s):

[Included]

[Inclu

# Race property of Lakedai. **Demographic and Other Baseline Characteristics**

# 7.4.1.1 Demographic and Other Baseline Characteristics

 $Min \le - \le 65, 65 < - \le 75,$ 

75 < - <= Max

[Male, Female]

[Hispanic or Latino, Not Hispanic or

Latino, Not Reported]

[White, Black or African American,

Native Hawaiian or Other Pacific

Islander, Asian (Asian Indian), Asian

(Chinese), Asian (Japanese), Asian (Korean), Asian (Other), Asian (Not

Reported), American Indian or

Alaska Native, Not Reported, Other]

Dose at Study Entry (months)

ISS Stage at Initial Diagnosis [I, II, III, Unknown]

**Patient Population Categories** [Relapsed Patients,

Refractory Patients,

le Lekins of Use Refractory and Relapsed Patients]

Type of Myeloma at Initial Diagnosis

**IgG** [Kappa, Lambda, Biclonal,

Unknown]

[Kappa, Lambda, Biclonal, ] **IgA** 

Unknown]

[Kappa, Lambda, Biclonal, IgD

Unknown]

IgE [Kappa, Lambda, Biclonal,

Unknown \

[Kappa, Lambda, Biclonal, **IgM** 

Unknown]

**Biclonal** Kappa, Lambda, Biclonal,

Unknown]

[Kappa, Lambda, Biclonal, Unknown

Unknown]

Other [Kappa, Lambda, Biclonal,

Unknown]

Durie-Salmon Stage at Initial [IA, IB, IIA, IIB, IIIA, IIIB,

Diagnosis Unknown] Lines of Prior Therapy [1, 2, 3]

Evidence of Lytic Bone Disease at [Yes, No, Unknown]

**Initial Diagnosis** 

Evidence of Extramedullary Disease [Yes, No, Unknown]

at Initial Diagnosis


Patients with a Bone Marrow

Transplant or Stem Cell Transplant

Type of Transplant Procedure [Allogenic, Autologous, Both,

Unknown]

Time Since Last Transplant to First

Dose at Study Entry (months)

Type of Prior Regimens [Velcade Contained,

Thalidomide Contained,

Thalidomide Refractory,

Lenalidomide Contained,

icable Terms of Use Corticosteroids Contained.

Dexamethasone,

Prednisone.

Other,

Carfilzomib Contained,

Melphalan Contained,

Other]

Type of Last Prior Regimen

[Velcade Contained,

Thalidomide Contained,

Thalidomide Refractory,

Lenalidomide Contained,

Corticosteroids Contained,

Dexamethasone,

Prednisone,

Other.

Carfilzomib Contained,

Melphalan Contained,

Other]

Patient was Relapsed on Last Prior

Therapy

Patient was Refractory on Last Prior

[Yes, No]

[Yes, No]

Therapy

Time Since Last Dose of Prior

Therapy to First Dose at Study Entry

(months)


Best Response to Prior Therapy

[Complete Response, Partial

Response, Stable Disease,

Progressive Disease, Unable to

Assess, Unknown]

Time Since Disease Progression on

Prior Therapy to First Dose at Study

Entry (months)

Patients with Prior Radiation

Time Since Last Prior Radiation to

First Dose at Study Entry (months)

Patients with Prior Surgery or Non-

**Radiation Procedures** 

Time Since Last Prior Surgery or Non-Radiation Procedure to First

Dose at Study Entry (months)

Prior IMiD Therapy [Exposed,

Thalidomide, Lenalidomide, Pomalidomide,

Naive]

[Yes, No]

Patient was Refractory to Any Prior

IMiD Therapy

Prior Proteasome Inhibitor Therapy [Exposed

Velcade,

Carfilzomib,

Naive]

Patient was Refractory to Any Prior [Yes, No]

Proteasome Inhibitor Therapy

Primary Refractory Patients [Progression Disease, Stable Disease]

ISS Stage for Myeloma at Study [I, II, III]

Entry

Evidence of Lytic Bone Disease [Present, Absent, Unknown]

Extramedullary Disease at Study [Yes, No, Unknown]

Entry

Serum M-Protein (g/L)

Urine M-Protein (g/24h)

Serum Creatinine (mg/dL) [Min $\leq$  -  $\leq$ 2, 2 $\leq$  -  $\leq$ Max]

Serum Albumin (g/L)  $[Min \le - <35, 35 \le - \le Max]$ 

 $\beta_2$ -microglobulin (mg/L) [Min<= - <3.5, 3.5<= - <5.5,

 $5.5 \le - \le Max$ 

Creatinine Clearance (mL/min)  $[Min \le -30, 30 \le -60,$ 

 $60 \le -490, 90 \le -4 \le Max$ 

Corrected Calcium (mmol/L)

Baseline ECOG Performance Status [0, 1, 2, 3, 4]

Baseline Hemoglobin (g/L)

Analytical


Method(s): (1) Summary of Demographics and Baseline Characteristics

icable reins of Use applicable applicable applicable to the applic Frequency distributions for categorical variables and descriptive statistics for

continuous variables will be provided.

7.4.1.2 Baseline Bone Marrow Evaluation and Extramedullary Disease Assessment

Full Analysis Set Analysis Set:

Analysis


Variable(s): Bone Marrow Aspiration

Number of Patients with Bone

Marrow Aspiration

Number of Patients with Adequate

Sample for Interpretation

% Plasma Cells [Available, Unable to Detect,

Not Available]

Bone Marrow Biopsy

Number of Patients with Bone

Marrow Biopsy

Number of Patients with Adequate

Sample for Interpretation

% Plasma Cells [Available, Unable to Detect,

Not Available]

% Marrow Cellularity [Available, Not Available]

Marrow Cellularity Status [Hypocellular, Hypercellular,

Normocellular, Unable to Assess]

Ommunohistochemistry or

Immunofluorescence for

Kappa/Lambda Ratio Performed

[Yes, No, Not Applicable]

Ratio Determined by Analysis of a

Minimum of 100 Plasma Cells

[Yes, No, Not Applicable]

% Plasma Cells in Bone Marrow

Kappa/Lambda Ratio

Bone Marrow Cytogenetic Results

Sample Collected? [Yes, No, Not Applicable]

Method of Assessment [Conventional/Karotype,

Molecular/FISH, Both]

Cytogenetic Results

(Conventional/Karotype) [Normal, Abnormal, Indeterminate]

Cytogenetic Results

e Terms of Use (Molecular/FISH) [Normal, Abnormal, Indeterminate]

Abnormality of Chromosomal

Aberrations

Subjects with Any Chromosomal [Del 13 or -13q, Del 17 or -17p]

Abnormalities t(4;14), t(6;14), t(8;14), t(11;14),

t(12;14), t(14;16), t(14;20), Hyperdiploidy, Hypodiploidy,

Non-hyperdiploidy,

1q amplification, 1q deletion, Other]

Cytogenetic Results [High Risk, Standard, Not Available]

Skeletal Survey

Result Within Normal Limits, Abnormal]

Lytic Bone Lesions Present [Yes, No, Indeterminate]

Imaging (Computed Tomography)

Result [Within Normal Limits, Abnormal]

Plasmacytomas Present [Yes, No, Indeterminate]

Imaging (Magnetic Resonance

Imaging)

Result [Within Normal Limits, Abnormal]

Plasmacytomas Present [Yes, No, Indeterminate]

Imaging (Positron Emission

Tomography)

PET Activity [FDG Positive, FDG Negative,

Indeterminate]

Property of Takeda. Fo Subjects with Plasmacytomas [Liver (Visceral), Lung (Visceral),

Node, Soft Tissue, Lytic Bone,

Other]

Number of Plasmacytomas

[1, 2, >=3]

Soft Tissue Plasmacytomas Total

Size (cm<sup>2</sup>)

Lytic Bone Plasmacytomas Total

Size (cm<sup>2</sup>)

Analytical

Method(s): (1) Baseline Bone Marrow Evaluation and Extramedullary Disease Assessment

licable terms of Use Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided.

### 7.4.1.3 Baseline Bone Marrow Cytogenetic Results

Analysis Set: Full Analysis Set

Analysis

[Del 13, Del 17, t(4;14), t(14;16), 1q Variable(s): Cytogenetics

amplification amplification

Analytical

Frequency distributions will be provided by the laboratory (central Method(s):

laboratory, local lab and total).

# 7.4.1.4 Disease Specific History – IMiD and Proteasome Inhibitor

Analysis Set: Full Analysis Set

Analysis

Exposed to Prior IMiD Therapy Variable(s):

Lenalidomide

Lenalidomide Refractory

Best Response [CR, PR, SD, PD, Unable to Assess,

Unknown]

Thalidomide Refractory

Best Response [CR, PR, SD, PD, Unable to Assess,

Unknown]

Pomalidomide

Pomalidomide Refractory

Best Response [CR, PR, SD, PD, Unable to Assess,

Unknown]

Property of Fakeda. For not halidomide Thalidom Exposed to Prior Proteasome

Velcade

Velcade Refractory

Best Response [CR, PR, SD, PD, Unable to Assess,

Unknown]

Carfilzomib

Carfilzomib Refractory

Best Response [CR, PR, SD, PD, Unable to Assess, Unknown]

Analytical

Method(s):

(1) Disease Specific History – IMiD and Proteasome Inhibitor
Frequency distributions for categorical variables will be provided. For the
analysis variables "Exposed to Prior IMiD Therapy", "Lenalidomide",
"Thalidomide", "Pomalidomide", "Exposed to Prior Proteasome Inhibitor
Therapy", "Velcade", and "Carfilzomib", the denominators for the
percentages will be the number of subjects in FAS. For the analysis variables
"Lenalidomide Refractory", "Thalidomide Refractory", "Pomalidomide
Refractory", "Velcade Refractory", and "Carfilzomib Refractory", the
denominators for the percentages will be the number of subjects who were
exposed to the specified therapy (Lenalidomide, Thalidomide,
Pomalidomide, Velcade, or Carfilzomib). For the analysis variable "Best
Response", the denominators for the percentages will be the number of
subjects who were refractory to the specified therapy (Lenalidomide,
Thalidomide, Pomalidomide, Velcade, or Carfilzomib).

7.4.1.5 Summary of Baseline Measurable Status in Subjects with only Abnormal Baseline Free Light Chain

Analysis Set: Full Analysis Set

Analysis

Variable(s): Free Light Chains (no Heavy Chain)

Measureable

Measureable by FLC only

Non-measureable

Analytical

Method(s):

(1) Summary of Baseline Measurable Status in Subjects with only Abnormal Baseline Free Light Chain

Frequency distributions for categorical variables will be provided.

7.4.1.6 Summary of New Primary Malignancy

Analysis Set: Full Analysis Set

Analysis

Variable(s): Subjects with any New Primary

Malignancy

New Primary Malignancy Disease

Type (On Treatment) [Categories will be based on actual

data]

New Primary Malignancy Disease

Type (Follow-up) [Myelodysplastic syndrome,

Acute myeloid leukaemia or related

precursor neoplasm,

Precursor lymphoid neoplasm,

Mature B-cell neoplasm,

Mature T-cell and NK-cell neoplasm,

Hodgkin lymphoma, Solid Tumor,

Other]

Analytical

Method(s): (1) Summary of New Primary Malignancy

Frequency distributions will be provided. Summaries will be provided using the new primary malignancy disease type and its detailed categories, where

the detailed categories will be sorted alphabetically.

### 7.5 Medical History and Concurrent Medical Conditions

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Medical History

**Concurrent Medical Conditions** 

Analytical

Method(s): (1) Medical History by Verbatim Term

(2) Concurrent Medical Conditions by Verbatim Term

Frequency distributions will be provided.

Summary will be provided using verbatim terms. A subject with multiple occurrences of medical history within a verbatim term will be counted only

once in that verbatim term.

### 7.6 **Medication History and Concomitant Medications**

Analysis Set: Safety Analysis Set

Analysis

Variable(s): **Concomitant Medications** 

Analytical

(1) Concomitant Medications by ATC Pharmacological Subgroup and WHO Method(s):

Generic Term

Frequency distributions will be provided. Concomitant medications are defined as medications with start dates occurring on or after date of first dose and before date of last dose + 30 days. WHO Drug dictionary will be used for coding. Summaries will be provided using ATC pharmacological subgroup and WHO generic term. ATC pharmacological subgroup will be sorted alphabetically and WHO generic term will be sorted in decreasing frequency based on the number of reports. A subject who has been administered several medications with the same WHO generic term will be counted only once for that WHO generic term.

### 7.7 Study Drug Exposure and Compliance

# Study Drug Exposure and Compliance

Analysis Set: Safety Analysis Set

Analysis

Total Amount of Doses Taken (mg) Property of Takeda Variable(s):

Total Number of Doses Taken

Number of Treated Cycles [>=1, >=2, >=3, >=4, >=5, >=6, >=7,

>=8, >=9, >=10, >=11, >=12, >=13,

>=14, >=15, >=16, >=17, >=18,

>=19, >=20, >=21, >=22, >=23,

>=24]

[Min<= - <50, 50<= - <80, Relative Dose Intensity (%)

 $80 \le -100, 100, 100 \le -100$ 

[1<= - <=3, 4<= - <=6, 7<= -<=9. Extent of Exposure (cycles)

10<= - <= 12, 13<= - <= 15,

Extent of Exposure (days)

Percent Drug Compliance (%)  $[Min \le - <50, 50 \le - <=65,$ 65< - <=80, 80< - <=100,

$$100 < - <= Max$$

# Analytical

Method(s): (1) Study Drug Exposure and Compliance – Ixazomib

(2) Study Drug Exposure and Compliance – Lenalidomide

(3) Study Drug Exposure and Compliance – Dexamethasone

(4) Study Drug Exposure and Compliance – Combination (Ixazomib, Lenalidomide, Dexamethasone)

Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided. For (4), only the number of treated cycles, extent of exposure (cycles), and extent of exposure (days) will be provided.

Mean and 95% CI plots of changes over time will be provided for the relative dose intensity. A treated cycle is defined as a cycle in which the patients received any amount of Ixazomib for (1), Lenalidomide for (2),

Dexamethasone for (3), and any of Ixazomib, Lenalidomide, Dexamethasone for (4).

# 7.7.1.2 Dose Modifications

Safety Analysis Set Analysis Set:

Analysis

Property of Takes Variable(s): Dose Modification

Cycle Delayed

Action on Drug [No Action Taken, Reduced

> Prescribed, Reduced Non-Prescribed, Increased Prescribed, Increased non-Prescribed, Held, Missed, Delayed,

Discontinued Permanently]

Number of Subjects with at least 1 Dose Reduction Number of Subjects with at least 2 Dose Reduction

Analytical

Method(s):

- (1) Dose Modifications Ixazomib
- (2) Dose Modifications Lenalidomide
- (3) Dose Modifications Dexamethasone

ins of Use Frequency distributions will be provided for overall, for every cycle from Cycle 1 to 18, and for Cycles 1-6, 7-12, 13-18, 19-21, 22-24, >=25. The analysis variable "dose modification" includes reduced prescribed, reduced non-prescribed, increased prescribed, increased non-prescribed, delayed, and discontinued permanently. For the analysis variable "Action on Drug", a subject will be counted once for each unique reason for dose modification that they have had over the course of the study. For "Action on Drug", the numerators for the percentages are the number of subjects with a dosing modification and the denominators are the total number of subjects with non-Property of Takeda. For non-commercial use only and missing dosing data. Dose reduction is defined as a prescribed reduction in dose over consecutive scheduled dosing days.

### **7.8 Efficacy Analysis**

### 7.8.1 **Primary Efficacy Endpoint(s)**

### 7.8.1.1 Primary Analysis

Analysis Set:

Analysis

Variable(s):

Analytical

Method(s):

VGPR
Overall Response (CR+PR (including sCR and VGPR))
VGPR or better (CR+VGPR)
SD
'D

1e VGPR or better (ervals w''' intervals will be provided in the response-evaluable analysis set as the primary analysis. The response rate and the 2-sided 95% confidence intervals will be provided for each analysis variable based on the confirmed best response.

The response rates and the 2-sided 95% confidence intervals will also be summarized based on the unconfirmed best response and the best response (confirmed or unconfirmed) at the end of each cycle (from Cycle 1 to Cycle 24).

The ORR is defined as the proportion of patients who achieved PR or better. Stacked bar graph will be provided for ORR (confirmed or unconfirmed) and ORR (confirmed) at the end of each cycle and overall.

### Sensitivity Analysis

Full Analysis Set

Analysis

Variable(s): CR

**sCR** 

PR

**VGPR** 

Kerms of Use

Overall Response (CR+PR (including sCR and VGPR))

VGPR or better (CR + VGPR)

SD

PD

Not Evaluable

Analytical

Method(s):

To check the robustness of the results, the same analyses as those in Section 7.8.1.1 will be performed using FAS, except for the summary based on the best response (confirmed or unconfirmed) at the end of each cycle and the stacked bar graphs for ORR. Non-evaluable subjects in FAS will only be included in the denominator when calculating the response rates. The VGPR or better (CR + VGPR) rate and the 2-sided 95% confidence intervals will be provided in FAS as the sensitivity analysis for the primary analysis. Non-evaluable subjects in FAS will be included in the analysis as Use only and not VGPR or CR.

# **Secondary Efficacy Endpoint(s)**

7.8.2.1 Progression-free Survival

Full Analysis Set Analysis Set:

**Analysis** 

Variable(s):

Analytical

Method(s):


For the PFS, the Kaplan-Meier curve [and the 25th, 50th (median), and 75th percentiles, if estimable] will be calculated with their 2-sided 95% CIs in FAS. Kaplan-Meier estimates will also be calculated at 6 months, 9 months, 12 months, 18 months, and 24 months with their 2-sided 95% CIs. The median follow-up time in months and its 2-sided 95% CI will also be provided.

PFS is defined as the time from the date of first study drug administration to the date of first documentation of PD or death from any cause, whichever occurs first. The number of subjects with events and the number of subjects censored will be provided as well as the reason for censoring. Patients without documentation of PD will be censored at the date of the last response assessment that is SD or better. The details regarding the handling of missing assessments and censoring are presented in the table below.

| Situation | Date of Progression | Outcome |
|---|---|---|
| Situation | or Censoring | Outcome |
| N 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | | C 1 |
| No baseline and/or no post baseline | Date of first dose | Censored |
| assessment, no subsequent | | ~~ |
| anticancer therapy after study | | Ne |
| treatment, no death | | · Cal |
| Disease progression documented | Date of next | Progressed |
| between scheduled visits | scheduled visit | |
| No documented death or disease | Date of last adequate | Censored |
| progression | assessment <sup>1</sup> | |
| Lost to follow-up, withdraw | Date of last adequate | Censored |
| consent before any documented | assessment <sup>1</sup> | |
| death or disease progression | 250 | |
| Death or progression after more | Date of last adequate | Censored |
| than 1 missed visit <sup>2</sup> | assessment <sup>1</sup> | |
| Alternate antineoplastic therapy | Date of last adequate | Censored |
| started prior to disease progression | assessment prior to | |
| | starting alternate | |
| , Cio | antineoplastic therapy | |
| Death before first post baseline | Date of death | Progressed |
| assessment | | |
| Death between adequate assessment | Date of death | Progressed |
| visits | | |

Adequate disease assessment is defined as there is sufficient data to evaluate a subject's disease status.

<sup>2</sup>: Death or progression occurs more than 90 days from previous adequate assessment.

# 7.8.2.2 Duration of Response

Analysis Set: Responders in the Full Analysis Set

Analysis

Variable(s): DOR

Analytical

Method(s): For the DOR, the Kaplan-Meier curve [and the 25<sup>th</sup>, 50<sup>th</sup> (median), and 75<sup>th</sup>

percentiles, if estimable will be calculated with their 2-sided 95% CIs for the

DOR is defined as the time from the date of first documentation of response to the first documentation of PD. Responders without documentation of PD. Will be censored at the date of their last response better. The number of a 1. censored will be provided as well as the reason for censoring. For the analysis of DOR, "response" will be defined as (1) VGPR or better Use only and subject (2) ORR (3) CR and the same analysis will be performed for each type of response.

### 7.8.2.3 Time to Progression

Full Analysis Set Analysis Set:

**Analysis** 

Variable(s): TTP

Analytical

Method(s):

Proberty of Lakeda.

For the TTP, the Kaplan-Meier curve [and the 25th, 50th (median), and 75th percentiles, if estimable] will be calculated with their 2-sided 95% CIs in FAS. Kaplan-Meier estimates will also be calculated at 6 months, 9 months, 12 months, 18 months, and 24 months with their 2-sided 95% CIs. TTP is defined as the time from the date of first study drug administration to the date of first documentation of PD. Patients without documentation of PD at the time of analysis will be censored at the date of their last response assessment that is SD or better. Patients with no response assessment will be censored at the first day of administration. Patients who do not experience progression and start new systemic therapy for multiple myeloma will be censored at the date of their last response assessment that is SD or better. The number of subjects with events and the number of subjects censored will be provided as well as the reason for censoring.

### 7.8.2.4 Overall Survival

Analysis Set: Full Analysis Set

Analysis

Variable(s): OS

Analytical

For the OS, the Kaplan-Meier curve [and the 25th, 50th (median), and 75th Method(s):

percentiles, if estimable] will be calculated with their 2-sided 95% CIs in FAS. Kaplan-Meier estimates will also be calculated at 6 months, 9 months, 12 months, 18 months, and 24 months with their 2-sided 95% CIs. The median follow-up time in months and its 2-sided 95% CI will also be

provided.

OS is defined as the time from the date of first study drug administration to the date of death. Subjects without documentation of death at the time of the analysis will be censored at the date when they were last known to be alive. The number of deaths and the number censored will be provided as well as

the reason for censoring.

# Additional Efficacy Endpoint(s)

### 7.8.3.1 Best M-Protein Response to Treatment

Response-evaluable Analysis Set Analysis Set:

Analysis

Best M-Protein Response Variable(s):

Property of Lakedai. For Response Category [100% Reduction, Categories:

Immunofixation Negative,

>=90% Reduction, >=50% Reduction]

[90 - <100% Reduction,

75 - <90% Reduction.

50 - <75% Reduction,

25 - <50% Reduction]

[<25% Reduction to <25% Increase,

>=25% Increase]

No Post-Baseline Assessment of Measurable M-Protein

Analytical

Method(s):

Frequency distribution will be provided. For subjects with measurable serum M-protein at baseline, the best M-protein response is the percent change from baseline to best (lowest) value post-baseline in serum M-protein. For subjects with non-measurable serum M-protein, but measurable urine M-protein, the best M-protein response is the percent change from baseline to best (lowest)? value post-baseline in urine M-protein. Mean and standard deviation plots of changes over time of serum M-protein will be provided for observed values and percent changes from baseline. A waterfall plot of serum M-protein will in the off be provided for the percent changes from baseline.

# 7.8.3.2 Time to Response

Responders in the Response-evaluable Analysis Set only and sulp Analysis Set:

Full Analysis Set

Analysis

VGPR or better (CR + VGPR) Variable(s):

Overall Response

Analytical

For the time to response, the Kaplan-Meier curve [and the 25<sup>th</sup>, 50<sup>th</sup> (median), Method(s):

and 75<sup>th</sup> percentiles, if estimable] will be calculated with their 2-sided 95% CIs, showing as cumulative distribution function. Kaplan-Meier estimates will also be calculated at 6 months, 9 months, 12 months, 18 months, and 24

months with their 2-sided 95% CIs.

Time to response is defined as the time from the date of first study drug administration to the date of first documentation of the confirmed response indicated in the analysis variable. Responders are defined as subjects with documentation of a confirmed response of the analysis variable. The number of subjects with events and the number of subjects censored will be provided.

The same analyses will be performed using FAS.

# 7.8.3.3 Duration of Follow-up

Analysis Set: Full Analysis Set

**Analysis** 

Variable(s): Duration of Follow-up

Analytical

For the duration of follow-up, the Kaplan-Meier estimates [the 25<sup>th</sup>, 50<sup>th</sup> Method(s):

(median), and 75<sup>th</sup> percentiles, if estimable] will be calculated with their 2-sided 95% CIs. Kaplan-Meier estimates of the follow-up rate will also be calculated at 6 months, 9 months, 12 months, 18 months, and 24 months with their 2-sided 95% CIs. The median follow-up time in months and its 2-sided 95% CI will also be provided.

Duration of follow-up is defined as time from the date of first study drug administration to the date of death or last known visit. The number of subjects with events and the number of subjects censored will be provided as well as the reason for censoring.

### 7.8.4 Statistical/Analytical Issues

7.8.4.1 Adjustments for Covariates

Not applicable.

7.8.4.2 Handling of Dropouts or Missing Data

Censoring rules have been described in each applicable section. For M-protein, values below the lower limit of quantification will be treated as zero.

7.8.4.3 Multicenter Studies

Treatment-by-center interaction will not be explored since this study is a single-arm study.

7.8.4.4 Multiple Comparison/Multiplicity

Not applicable.

7.8.4.5 Use of an "Efficacy Subset" of Subjects

In addition to analyses on the primary endpoint using the response-evaluable analysis set, a secondary analysis will also be performed using the FAS to examine the robustness of the results.

7.8.4.6 Active-Control Studies Intended to Show Equivalence or Non-Inferiority Not applicable.

7.8.4.7 Examination of Subgroups

Analysis Set: Response-evaluable Analysis Set

Full Analysis Set

Analysis

Variable(s): CR

**sCR** 

PR

**VGPR** 

Overall Response (CR+PR (including sCR and VGPR))

VGPR or better (CR + VGPR)

SD

PD

Subgroup(s): Age (years)

Sex

[Min<= - <=65, 65< - <=75, 100 75< - <=Max] Male, Female] High Risk !!' Cytogenetic Risk

t(14;16)}, Non-High Risk]

ISS Stage for Myeloma at Study [I, II, III]

Entry

Lines of Prior Therapy [1, 2 or 3]

Prior Proteasome Inhibitor Therapy [Exposed, Naive] [Exposed, Naive] Prior IMiD Therapy

Thalidomide Refractory [Yes, No] Refractory to Any Line of Prior [Yes, No]

Therapy

Patient was Refractory on Last Prior [Yes, No]

Therapy

Relapsed and/or Refractory [Relapsed, Refractory, Relapsed and

Refractory]

Prior Velcade Therapy [Exposed, Naive]

Creatinine Clearance (mL/min)  $[Min \le - <60, 60 \le - <=Max]$ 

Baseline ECOG Performance Status [0 or 1, 2]

Prior Lenalidomide Therapy [Exposed, Naive] Prior Thalidomide Therapy [Exposed, Naive]

Method(s): The same analyses as those in Sections 7.8.1.1 and 7.8.1.2 will be performed

> with the confirmed best response for each subgroup. A forest plot will be produced using the VGPR or better (CR+VGPR) rate and the 2-sided 95%

confidence intervals.

### 7.8.4.8 Examination of Subgroups – Summary Table

Analysis Set: Response-evaluable Analysis Set

Full Analysis Set

Analysis

Variable(s): ORR

> VGPR or better CR or better

Subgroup(s): Age (years)

Sex

Cytogenetic Risk

[Min<= - <=65, 65< - <=75, 75< - <=Max] Male, Female] Not Availab' igh r High Risk, High Risk (del17), High Risk t(4;14), High Risk t(14;16)]

Baseline ECOG Performance Status

Prior Lines of Therapy per Takeda

review with SCT, without SCT,

[0, 1, 2]

with SCT, without SCT,

3,

with SCT, without SCT]

Relapsed/Refractory Type [Relapsed, Refractory,

Relapsed and Refractory,

Primary Refractory]

Prior Proteasome Inhibitor [Exposed, Naive,

Refractory (Takeda),

Vc-Refractory (Takeda),

CFZ-Refractory (Takeda)]

Prior IMiD [Exposed, Naive,

Refractory (Takeda),

Thal-Refractory (Takeda), Len-Refractory (Takeda)]

ISS stage at Study Entry [I, II, III]

Property of Takedai. For Best Response [>=CR, >=VGPR, >=PR, SD, PD]

Creatinine Clearance (mL/min)  $[Min \le - <60, 60 \le - <=Max]$ 

1 Prior Line with SCT

High Risk

ISS 3

., Naive]
[Yes, No]
[0<= - <12, 12<= - <24, 24<= - <36,
36<= - <= Max]
[Exposed, Naive]

Single S Prior IMiD Thalidomide Lenalidomide

Maintenance Therapy (Takeda)

Time from Last SCT to First Dose

(Months) Prior PI

1 Prior Line with SCT

Single vs. Double SCT [Single SCT, Double SCT]

With Velcade + Thalidomide [Yes, No] With Velcade + Lenalidomide

[CR, PR, SD or PD] Best Response on Prior SCT

**ECOG** 

Low Bone Marrow Cellularity [Yes, No, Missing] Cytogenetic Risk [Not Available,

1 Line with SCT, Others]

Analytical

Frequency distributions for each analysis variable will be provided for each Method(s):

subgroup.

### Pharmacokinetic/Pharmacodynamic Analysis 7.9

### Pharmacokinetic Analysis

Not applicable.

### Pharmacodynamic Analysis

Not applicable. Not applicable.

### Other Outcomes
## **Safety Analysis** 7.11

# 7.11.1 Adverse Events

7.11.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set:

Analysis

Variable(s):

Analytical

Property of Takedai.

Method(s):

- The following summaries will be provided.

  (1) Overview of Treatment-Emergent Adverse Events

  1) Any adverse event

  2) Grade 3 or higher adverse event

  3) Drug-related adverse event

  4) Drug-related grade 3 or '

  5) Serious adver

  6) Dru

  - 6) Drug-related serious adverse event
  - 7) Adverse events resulting in any study drug dose reduction
  - 8) Adverse events resulting in any study drug dose modification
  - Adverse events resulting in any study drug discontinuation
  - 10) On-study deaths

For summary 8), dose modification will include dose reduction, dose increase, dose delay, and dose discontinuation.

TEAEs will be counted according to the rules below.

# Number of subjects

Summaries for 3), 4), and 6)

A subject with occurrences of TEAE in both categories (i.e., Related and Not Related) will be counted once in the Related category.

Summaries for 2) and 4)

A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.

• Summaries other than 2), 3), 4), and 6) A subject with multiple occurrences of TEAE will be counted only once.

# 7.11.1.2 Overview of Treatment-Emergent Adverse Events by Subgroups

Analysis Set: Safety Analysis Set

Analysis

Variable(s): TEAE

Subgroup(s): Cycles [1-6, 7-12, 13-18, >=19]

Sex [Male, Female]

Creatinine Clearance (mL/min) [Min<= - <60, 60<= - <=Max]

Analytical

Method(s): The same overview summary as Section 7.11.1.1 will be provided for each subgroup category.

(1) Overview of Treatment-Emergent Adverse Events by Cycle in Subjects with >= 12 Cycles Exposure

(2) Overview of Treatment-Emergent Adverse Events by Sex

(3) Overview of Treatment-Emergent Adverse Events by Creatinine Clearance

The summary in (1) will be based on subjects who have completed 12 cycles or more of the study drug.

# 7.11.1.3 Displays of Treatment-Emergent Adverse events

Analysis Set: Safety Analysis Set

Analysis

Variable(s): TEAE

Categories: Intensity [Grade 1, Grade 2, Grade 3, Grade 4,

Grade 5]

Time of Onset (Cycle) [1-3, 4-6, 7-9, 10-12, 13-15,

16 - 18, 19 - 21, 22 - 24

Analytical

Method(s): The following summaries will be provided using frequency distribution.

TEAEs will be coded using the MedDRA and will be summarized using

SOC, HLT, and PT.

SOC, HLT, and PT will be sorted in decreasing frequency for tables provided by SOC, HLT, and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. PT will be sorted in decreasing frequency for tables provided by PT only.

(1) Treatment-Emergent Adverse Events by System Organ Class, High


- Level Term, and Preferred Term
- (2) Treatment-Emergent Adverse Events by Preferred Term
- (erms of Use (3) Treatment-Emergent Drug-Related Adverse Events by System Organ Class, High Level Term, and Preferred Term
- (4) Treatment-Emergent Grade 3 or Higher Adverse Events by System Organ Class, High Level Term, and Preferred Term
- (5) Treatment-Emergent Grade 3 or Higher Adverse Events by Preferred Term
- (6) Treatment-Emergent Drug-Related Grade 3 or Higher Adverse Events by System Organ Class, High Level Term, and Preferred Term
- (7) Treatment-Emergent Grade 4 Adverse Events by System Organ Class, High Level Term, and Preferred Term
- (8) Intensity of Treatment-Emergent Adverse Events by System Organ Class, High Level Term, and Preferred Term
- (9) Intensity of Treatment-Emergent Drug-Related Adverse Events by System Organ Class, High Level Term, and Preferred Term
- (10) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class, High Level Term, and Preferred Term
- (11) Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term, and Preferred Term
- (12) Treatment-Emergent Drug-Related Serious Adverse Events by System Organ Class, High Level Term, and Preferred Term
- (13) Treatment-Emergent Adverse Events by System Organ Class, High Level Term, and Preferred Term Over Time
- (14) Most Frequent Non Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (15) Summary of Treatment-Emergent Adverse Events which Resulted in Dose Reduction by System Organ Class and Preferred Term
- (16) Summary of Treatment-Emergent Adverse Events which Resulted in Dose Held by System Organ Class and Preferred Term
- (17) Summary of Treatment-Emergent Adverse Events which Resulted in Dose Discontinuation by System Organ Class and Preferred Term The frequency distribution will be provided according to the rules below. Number of subjects
- Summary tables other than (4) to (9) and (13)

Probeity of Lakeda.

A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within an HLT will be counted only once in that HLT. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the safety analysis set.

Summary tables for (4) to (9)
 A subject with multiple occurrences of TEAE within a SOC, an HLT, or a PT will be counted only once for the TEAE with the maximum intensity.
 Percentages will be based on the number of subjects in the safety analysis

• Summary table for (13)

Dexamethasone.

A subject with a TEAE that occurs in more than one interval is counted in all the intervals that the TEAE occurs. For each time interval, a subject with multiple occurrences of TEAE within a SOC, an HLT, or a PT will be counted only once in that SQC, HLT, or PT.

When calculating percentages for each time interval, the number of subjects at risk (i.e., subjects who either have an exposure or have an occurrence of TEAE, during or after the corresponding time interval) will be used as the denominator. The number of subjects whose onset of any one of the TEAEs is within the time interval will be used as the numerator.

- Summary table for (14)
   Most frequent non-serious TEAEs refer to PTs that are not serious whose percentages are at least 5%.
- Summary table for (15)
  TEAEs which resulted in dose reduction in Ixazomib, in Lenalidomide,
  and in Dexamethasone will each be displayed, as well as the TEAEs which
  resulted in dose reduction in any of Ixazomib, Lenalidomide, or
- Summary table for (16)
  TEAEs which resulted in dose held in Ixazomib, in Lenalidomide, and in Dexamethasone will each be displayed, as well as the TEAEs which resulted in dose held in any of Ixazomib, Lenalidomide, or Dexamethasone.
- Summary table for (17)

  TEAEs which resulted in dose discontinuation in Ixazomib, in

  CONFIDENTIAL

Lenalidomide, and in Dexamethasone will each be displayed.

licable Terms of Use 7.11.1.4 Displays of Treatment-Emergent Adverse Events of Clinical Importance and Haemorrhage

Analysis Set: Safety Analysis Set

Analysis

Variable(s): TEAE of clinical importance

Treatment-emergent haemorrhage adverse events

[Grade 1, Grade 2, Grade 3, Grade 4, Grade 5] NCI CTCAE Grade Categories:

Analytical

Adverse events of clinical importance will include diarrhea, rash, Method(s):

> neutropenia, thrombocytopenia, nausea, peripheral neuropathy, vomiting, arrhythmias, renal, liver impairment, hypotension, heart failure, new primary malignancy, myocardial infarction, and encephalopathy. The following summaries will be provided using frequency distribution. For (2) and (3), descriptive statistics will be provided. For (3), time to resolution from the first onset of the AE will be summarized. If no date of resolution is recorded, then the last date of visit will be used as the date of resolution.

> TEAEs will be coded using the MedDRA and will be summarized using PT for (1) to (6). For (1), PT will be sorted in decreasing frequency. For (4) to (6), AECI and PT will both be sorted alphabetically. A subject with multiple occurrences of TEAE within a PT will be counted only once for the TEAE with the maximum intensity. For (4), TEAEs of clinical importance which resulted in dose reduction in Ixazomib, in Lenalidomide, and in Dexamethasone will each be displayed, as well as TEAEs of clinical

importance which resulted in dose reduction in any of Ixazomib, Lenalidomide, or Dexamethasone. For (5), TEAEs of clinical importance which resulted in dose held in Ixazomib, in Lenalidomide, and in Dexamethasone will each be displayed, as well as TEAEs of clinical importance which resulted in dose held in any of Ixazomib, Lenalidomide, or Dexamethasone. For (6), TEAEs of clinical importance which resulted in dose discontinuation in Ixazomib, in Lenalidomide, and in Dexamethasone will each be displayed, as well as TEAEs of clinical importance which resulted in dose discontinuation in any of Ixazomib, Lenalidomide, or

Dexamethasone. For (7), TEAEs will be summarized using SOC, HLT, and

PT, where SOC, HLT, and PT will be sorted in decreasing frequency. TEAEs will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (Version 4.03).

- (1) Treatment-Emergent Adverse Events of Clinical Importance by Preferred Term and NCI CTCAE Grade
- (2) Summary of Time to First Onset in Treatment-Emergent Adverse Events of Clinical Importance
- (3) Summary of Time to Resolution in Treatment-Emergent Adverse Events of Clinical Importance
- (4) Treatment-Emergent Adverse Events of Clinical Importance which Resulted in Dose Reduction by Preferred Term
- (5) Treatment-Emergent Adverse Events of Clinical Importance which Resulted in Dose Held by Preferred Term
- (6) Treatment-Emergent Adverse Events of Clinical Importance which Resulted in Dose Discontinuation by Preferred Term
- (7) Treatment-Emergent Haemorrhage Adverse Events by System Organ Class, High Level Term, and Preferred Term
- (8) Treatment-Emergent Adverse Events of Clinical Importance, Grades and Concomitant Medications by ATC Pharmacological Subgroup and WHO Generic Term

7.11.1.5 Summary of Treatment-Emergent Adverse Events Overall, and by Toxicity, Seriousness, Relatedness, Discontinuation, and Dose Modification

Analysis Set: Safety Analysis Set

Analysis

Variable(s): TEAE

TEAE of clinical importance

Analytical

Method(s):

The following summaries will be provided using frequency distribution. The summaries will include the number and percentages of subjects who had any TEAEs, drug-related TEAEs, Grade 3 or higher TEAEs, Grade 3 or higher drug-related TEAEs, serious TEAEs, TEAEs resulting in death, TEAEs leading to study drug discontinuation, TEAEs which resulted in dose reduction, dose held, and dose delayed in any of Ixazomib, Lenalidomide, or Dexamethasone. TEAEs will be coded using the MedDRA and will be

summarized using SOC and PT. SOC and PT will be sorted in decreasing frequency.

- (1) Summary of Treatment-Emergent Adverse Events Overall, and by Toxicity, Seriousness, Relatedness, Discontinuation, and Dose Modification
- (erms of Use (2) Summary of Treatment-Emergent Adverse Events of Clinical Importance ating applifect to the applif Overall, and by Toxicity, Seriousness, Relatedness, Discontinuation, and Dose Modification

# 7.11.2 Clinical Laboratory Evaluations

# 7.11.2.1 Hematology and Blood Chemistry

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Hematology

> Hematocrit Platelet Count Hemoglobin Neutrophils **WBC** Count Lymphocytes

Serum Chemistry

Blood Urea Nitrogen Creatinine Total Bilirubin

Uric Acid Alkaline Phosphatase Lactate dehydrogenase

(LDH)

**AST** ALT Albumin Potassium Glucose Sodium Chloride Carbon dioxide Magnesium

Calcium Phosphate Thyroid Stimulating

Hormone (TSH)

Categories: Intensity [Grade 0, Grade 1, Grade 2, Grade 3, Grade 4]

Hematology: Screening, Baseline, Cycle 1 Day 1, Cycle 1 Day 7, Cycle 1

Day 14, Cycle 1 Day 21, Cycle 2 Day 1, Cycle 2 Day 7, Cycle 2 Day 14,

Cycle 2 Day 21, Cycle 3 Day 1, Cycle 3 Day 14, Cycle 4 Day 1, Cycle 5 Day

1, Cycle 6 Day 1, ... (up to the maximum cycle), End of Treatment, Last

Assessment

Serum Chemistry: Screening, Baseline, Cycle 1 Day 1, Cycle 2 Day 1, Cycle

3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1, ... (up to the

maximum cycle), End of Treatment, Last Assessment

Analytical

Method(s): For each variable, (1) will be provided.

For applicable variables, (2), (3), and (4) will be provided.

NCI CTCAE (Version 4.03) will be used for grading. Last Assessment is defined as the last measurement prior to or on the last visit conducted 30 days after the last dose of study drug regimen.

Laboratory test results from the central laboratory will be used when they are available. Laboratory test results from local laboratory will be used only when no central laboratory test result exists at the same scheduled sample collection time point.

- (1) Summary of Laboratory Test Results and Change from Baseline by Visit Descriptive statistics for observed values for each visit and changes from baseline will be provided.
- (2) Case Plots
  Plots over time for each subject will be presented for platelet count.
- (3) Line Plot of Platelet Count Over Time

  For the platelet count, the overall median over time will be presented.
- (4) Maximum Grade Shift from Baseline of Laboratory Parameters

  The maximum (worst) post-baseline grade will be determined for each subject. Shift tables showing the number of subjects in each grade category at baseline and post-baseline visit will be provided using evaluable data.

# 7.11.3 Vital Signs and Weight

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Systolic Blood Pressure (mmHg)

Diastolic Blood Pressure (mmHg)

Heart Rate (bpm)

Respiratory Rate (bpm)

Temperature (C)

Weight (kg)

Visit: Screening, Baseline, Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1,

Cycle 4 Day 1, ... (up to the maximum cycle), End of Treatment,

Last Assessment

Analytical

ns of Use

Method(s): For each variable, the following summaries will be provided.

> Last Assessment is defined as the last measurement prior to or on the last visit conducted 30 days after the last dose of study drug regimen.

(1) Summary of Vital Signs Parameters and Change from Baseline by Visit and subject to the applicable and, 1.7 Descriptive statistics for observed values for each visit and changes from baseline will be provided.

## 7.11.4 12-Lead ECGs

Not applicable.

# 7.11.5 Other Observations Related to Safety

7.11.5.1 ECOG Performance Status

Analysis Set: Safety Analysis Set

Analysis

**ECOG Performance Status** Variable(s):

Categories: **ECOG Score** 

Screening, Baseline, Cycle 2 Day 1, Cycle 3 Day 1, ... (up to the maximum Visit:

cycle), End of Treatment, Dast Assessment

Analytical

For each variable, the following summaries will be provided. Method(s):

> Last Assessment is defined as the last measurement prior to or on the last visit conducted 30 days after the last dose of study drug regimen.

- (1) ECOG Performance Status Data Measured Over Time Descriptive statistics for observed values for each visit and changes from baseline will be provided.
- (2) ECOG Performance Score Shift from Baseline to Post-Baseline Assessments Over Time Shift tables showing the number of subjects in each ECOG score category at baseline and each post-baseline visit will be provided.

7.11.5.2 Subsequent Anti-Cancer Therapy

Safety Analysis Set

Variable(s): Subsequent Anti-Cancer Therapy

Analytical

Method(s): (1) Subsequent Anti-Cancer Therapy by Class of Agent and WHO Generic Term

Frequency distributions will be provided.

# 7.12 Interim Analysis

Analysis is planned to be performed twice during the study. The primary analysis is planned to be performed using the data obtained at approximately 12 months from the enrollment of the last patient. The final analysis is planned to be performed after the final database lock using the data obtained at approximately 24 months from the enrollment of the last patient. The timing of analysis may be changed or additional analysis may be added upon request of the regulatory authorities.

# 7.13 Changes in the Statistical Analysis Plan

The analyses in the statistical analysis plan do not differ from the analyses specified in the protocol.

Changes from the previous version of SAP are listed below.

# Page 20, Section 7.4.1.3 Baseline Bone Marrow Cytogenetic Results

# **Added Text**

Analysis Set: Full Analysis Set

Analysis

Variable(s): Cytogenetics [Del 13, Del 17, t(4;14), t(14;16), 1q

amplification]

Analytical

Method(s): Frequency distributions will be provided by the laboratory (central

laboratory, local lab and total).

## **Rationale for Amendment**

This section has been added.

# Page 22, Section 7.5 Medical History and Concurrent Medical Conditions

# **Existing Text**

(2) Concurrent Medical Conditions by <u>System Organ Class and Preferred Term</u> Frequency distributions will be provided.

For (1), summary will be provided using verbatim terms. A subject with multiple occurrences

occurrences of concurrent medical condition within a SOC will be counted only once in that SOC. A subject with multiple occurrences of concurrent medical condition within a PT will be counted only once in that PT.

Revised Text

(2) Concurrent Medical C.

Frequency distributions will be provided.

Summary will be provided using verbatim terms. A subject with multiple occurrences of medical history within a verbatim term will be counted only once in that verbatim term.

# **Rationale for Amendment**

Concurrent Medical Conditions has not been coded by MedDR

# Page 30, Section 7.8.3.1 Best M-Protein Response to Treatment

# **Existing Text**

Mean and standard deviation plots of changes over time will be provided for observed values and percent changes from baseline. A waterfall plot of will be provided for the percent changes from baseline.

## **Revised Text**

Mean and standard deviation plots of changes over time of serum M-protein will be provided for observed values and percent changes from baseline. A waterfall plot of serum M-protein will be provided for the percent changes from baseline.

# **Rationale for Amendment**

To clarify the analytical method.

# Page 31, Section 7.8.3.2 Time to Response

# **Existing Text**

For the time to response, the Kaplan-Meier curve [and the 25<sup>th</sup>, 50<sup>th</sup> (median), and 75<sup>th</sup> percentiles, if estimable will be calculated with their 2-sided 95% CIs.

# **Revised Text**

For the time to response, the Kaplan-Meier curve [and the 25<sup>th</sup>, 50<sup>th</sup> (median), and 75<sup>th</sup> percentiles, if estimable] will be calculated with their 2-sided 95% CIs, showing as cumulative distribution function.

## Rationale for Amendment

To clarify the analytical method.

# Page 31, Section 7.8.3.2 Time to Response

# **Existing Text**

The number of subjects with events and the number of subjects censored will be provided as well as the reason for censoring.

# **Revised Text**

The number of subjects with events and the number of subjects censored will be provided. ,ct to the appi

# **Rationale for Amendment**

To clarify the analytical method.

# Page 31, Section 7.8.3.3 Duration of Follow-up

# **Existing Text**

For the duration of follow-up, the Kaplan-Meier curve [and the 25<sup>th</sup>, 50<sup>th</sup> (median), and 75<sup>th</sup> percentiles, if estimable] will be calculated with their 2-sided 95% CIs. Kaplan-Meier estimates will also be calculated at 6 months, 9 months, 12 months, 18 months, and 24 months with their 2-sided 95% CIs.

# **Revised Text**

For the duration of follow-up, the Kaplan-Meier estimates [the 25th, 50th (median), and 75th percentiles, if estimable] will be calculated with their 2-sided 95% CIs. Kaplan-Meier estimates of the follow-up rate will also be calculated at 6 months, 9 months, 12 months, 18 months, and 24 months with their 2-sided 95% CIs.

# **Rationale for Amendment**

To clarify the analytical method.

# Page 32, Section 7.8.4.2 Handling of Dropouts or Missing Data

# Adding Text

For M-protein, values below the lower limit of quantification will be treated as zero.

# **Rationale for Amendment**

There have been the values "below the lower limit of quantification".

# Page 32, Section 7.8.4.7 Examination of Subgroups

# **Existing Text**

 $[Min \le - <60, 60 \le - <=Max]$ Creatinine Clearance (mL/min)

 $[Min \le - <50, 50 \le - <=Max]$ 

## **Revised Text**

Creatinine Clearance (mL/min)

 $[Min \le - <60, 60 \le - <=Max]$ 

# **Rationale for Amendment**

This subgroup has not been needed.

# Page 34, Section 7.8.4.8 Examination of Subgroups – Summary Table

**Existing Text** 

Prior Proteasome Inhibitor [Exposed, Naive,

Refractory,

Vc-Refractory (Takeda), CFZ-Refractory (Takeda)]

Prior IMiD [Exposed, Naive,

Refractory,

Thal-Refractory (Takeda), Len-Refractory (Takeda)]

**Revised Text** 

Prior Proteasome Inhibitor Exposed, Naive,

Refractory (Takeda),

Vc-Refractory (Takeda), CFZ-Refractory (Takeda)]

Prior IMiD [Exposed, Naive,

Refractory (Takeda),

Thal-Refractory (Takeda), Len-Refractory (Takeda)]

**Rationale for Amendment** 

To correct the miswritings.

# Page 34, Section 7.8.4.8 Examination of Subgroups – Summary Table

**Existing Text** 

Creatinine Clearance (mL/min) [Min<= - <50, 50<= - <=Max]

[Min<= - <50, 50<= - <60,

 $60 \le - \le Max$ 

[Min<= - <60, 60<= - <=Max]

**Revised Text** 

Creatinine Clearance (mL/min)  $[Min \le - \le 60, 60 \le - \le Max]$ 

**Rationale for Amendment** 

These subgroups have not been needed.

# Page 34, Section 7.8.4.8 Examination of Subgroups – Summary Table

# **Existing Text**

Maintenance Therapy [Yes, No]

Time from SCT to First Dose  $[0 \le -12, 12 \le -24, 24 \le -36,$ 

 $(Months) 36 \le - \le Max$ 

**Revised Text** 

Maintenance Therapy (<u>Takeda</u>) [Yes, No]

Time from <u>Last SCT</u> to First Dose  $[0 \le -12, 12 \le -24, 24 \le -36,$ 

 $(Months) 36 \le - \le Max$ 

**Rationale for Amendment** 

To clarify the analytical method.

# Page 37, Section 7.11.1.2 Overview of Treatment-Emergent Adverse Events by Subgroups

**Existing Text** 

Creatinine Clearance (mL/min) [Min <= - <30, 30 <= - <60,

 $60 \le -890, 90 \le -880$ 

**Revised Text** 

Creatinine Clearance (mL/min)  $[Min \le - <60, 60 \le - \le Max]$ 

**Rationale for Amendment** 

This subgroup has been changed.

# Page 40, Section 7.11.1.3 Displays of Treatment-Emergent Adverse events

# **Existing Text**

Summary table for (17)

TEAEs which resulted in dose discontinuation in Ixazomib, in Lenalidomide, and in Dexamethasone will each be displayed, as well as the TEAEs which resulted in dose discontinuation in any of Ixazomib, Lenalidomide, or Dexamethasone.

# **Revised Text**

Summary table for (17)

TEAEs which resulted in dose discontinuation in Ixazomib, in Lenalidomide, and in Dexamethasone will each be displayed.

# **Rationale for Amendment**

The deleted portion has been duplicated.

# Page 40, Section 7.11.1.4 Displays of Treatment-Emergent Adverse Events of Clinical Importance and Haemorrhage

# **Adding Text**

(9) Treatment-Emergent Adverse Events of Clinical Importance, Grades and Concomitant Medications by ATC Pharmacological Subgroup and WHO Page 43, Section 7.11.2.1 Hematology and Blood Chemistry

Existing Text

(2) Case Plots

Plots over time for Generic Term

Plots over time for each subject will be presented for platelet count and neutrophils.

# **Revised Text**

**(2)** Case Plots

Plots over time for each subject will be presented for platelet count.

# **Rationale for Amendment**

Property of Fakeda. For non-comme The case plot of neutrophils has not been needed.



# STATISTICAL ANALYSIS PLAN

**STUDY NUMBER: C16028** 

\*Policable Terms of Use A Phase 2, Open-Label, Multicenter Study of Ixazomib Plus Lenalidomide and Dexamethasone in Adult Japanese Patients With Relapsed and/or Refractory Multiple Myeloma

# PHASE 2

Version: 1

Date: 16 August 2017

Prepared by:

PPD PPD

Based on:

Protocol Version: Amendment 1 Protocol Date: 25 November 2016

## CONFIDENTIAL PROPERTY OF TAKEDA

This document is a confidential communication of Takeda. Acceptance of this document constitutes the agreement by the recipient that no information contained herein will be published or disclosed without written authorization from Takeda.

Property of The Bank of the Ba

# 2.0 TABLE OF CONTENTS

| 1.0 | TI | ITLE PAGE | 1 |
|---|---|---|---|
| | 1.1 | Approval Signatures | 2 |
| 2.0 | TA | ABLE OF CONTENTS | 3 |
| 3.0 | LI | ABLE OF CONTENTSIST OF ABBREVIATIONS | |
| 4.0 | OH | BJECTIVES | <i>2</i> 7 |
| | 4.1 | Primary Objectives Secondary Objectives Additional Objectives Study Design NALYSIS ENDPOINTS DETERMINATION OF SAMPLE SIZE METHODS OF ANALYSIS AND PRESENTATION | 7 |
| | 4.2 | Secondary Objectives | 7 |
| | 4.3 | Additional Objectives | 7 |
| | 4.4 | Study Design | 7 |
| 5.0 | Aì | NALYSIS ENDPOINTS | 9 |
| 6.0 | DE | ETERMINATION OF SAMPLE SIZE | 9 |
| 7.0 | M | METHODS OF ANALYSIS AND PRESENTATION | 10 |
| | 7.1 | General Principles | 10 |
| | 7.1 | .1.1 Study Definitions | 10 |
| | 7.1 | .1.2 Definition of Study Visit Windows | 11 |
| | 7.1 | .1.3 Significance Level and Confidence Coefficient | 11 |
| | 7.2 | Analysis Sets | 11 |
| | 7.3 | Disposition of Subjects | 12 |
| | 7.3 | .3.1 Study Information | 12 |
| | 7.3 | .3.2 Number of Subjects Who Entered the Treatment Period by Site | 12 |
| | 7.3 | .3.3 Disposition of Subjects | 12 |
| | 7.3 | .3.4 Protocol Deviations and Analysis Sets | 13 |
| | 7.4 | Demographic and Other Baseline Characteristics | 14 |
| | 7.5 | Medical History and Concurrent Medical Conditions | 22 |
| | 7.6 | Medication History and Concomitant Medications | 23 |
| | 7.7 | Study Drug Exposure and Compliance | 23 |
| | 7.8 | Efficacy Analysis | 26 |
| | 7.8 | 8.1 Primary Efficacy Endpoint(s) | 26 |
| / | 7.8 | .8.2 Secondary Efficacy Endpoint(s) | 27 |
| | 7.8 | .8.3 Additional Efficacy Endpoint(s) | 30 |
| ) | 7.8 | .8.4 Statistical/Analytical Issues | 32 |
| | 7.9 | Pharmacokinetic/Pharmacodynamic Analysis | 35 |
| | 7.9 | .9.1 Pharmacokinetic Analysis | 35 |
| | 7.9 | .9.2 Pharmacodynamic Analysis | 35 |
| | 7.10 | Other Outcomes | 35 |
| | 7.11 | Safety Analysis | 36 |
| | 7 1 | 11.1 Adverse Events | 36 |

## 3.0 LIST OF ABBREVIATIONS

5-HT3

ADL

ΑE

anization
graphy
alon
deoxyribonucleic acid
duration of response
Eastern Cooperative Oncology Group
electronic case report form
and of Treatment (visit)
ill analysis set
nale patients of childbesited States Food
rescent in Fight ALT **ANC** AST **BUN** 

CBC CI  $CO_2$ CR

**CRO** 

CT**CYP** 

Del

**DNA** DOR

**ECOG** 

eCRF **EOT FAS** 

**FCBP FDA** 

**FISH** 

free light chain **FLC** Good Clinical Practice **GCP** 

granulocyte colony stimulating factor G-CSF

**GVHD** graft-versus-host disease **HBcAb** hepatitis B core antibody

**HBV** hepatitis B virus ъ ICH IMir **HCV** hepatitis C virus

human immunodeficiency virus

Investigator's Brochure

International Conference on Harmonisation

immunomodulatory drugs

**IMWG** International Myeloma Working Group

IRB institutional review board **ISS** international staging system

IUD intrauterine device

IV intravenous; intravenously lenalidomide and dexamethasone LenDex

LDH lactate dehydrogenase

MedDRA Medical Dictionary for Regulatory Activities **MHRA** Medicines and Healthcare products Regulatory Agency

MM multiple myeloma

MRI magnetic resonance imaging

NCI CTCAE National Cancer Institute Common Terminology Criteria for Adverse Events

**NDMM** newly diagnosed multiple myeloma

ORR overall response rate OS overall survival

PD progressive disease (disease progression)

PET positron emission tomography **PFS** progression-free survival

**PMDA** Pharmaceuticals and Medical Devices Agency **PML** progressive multifocal leukoencephalopathy

applicable Terms of Use progressive municipal reukoencephalopathy polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin **POEMS** 

changes

PR partial response

**PRES** posterior reversible encephalopathy syndrome.

PTE pretreatment event RNA ribonucleic acid

relapsed and/or refractory multiple myeloma **RRMM** 

SAE serious adverse event SAP statistical analysis plan sCR stringent complete response

stable disease SD

**SPEP** serum protein electrophoresis

**SUSAR** suspected unexpected serious adverse reaction

treatment-emergent adverse event **TEAE** TEN toxic epidermal necrolysis

time to first occurrence of maximum (peak) concentration  $T_{\text{max}}$ 

**TSH** thyroid stimulating hormone

TTP time to progression

ULN upper limit of the normal range urine protein electrophoresis very good partial response

white blood cell

World Health Organization

## 4.0 **OBJECTIVES**

10 determine VGPR or better (VGPR + CR) rate in response-evaluable analysis set\*

\*Defined as patients who received at least one dose of ixazomib and had measurable disease at baseline, and at least one post baseline response assessment.

4.2 Secondary Objectives

• To determine progression-free survival (PFS)

• To determine overall response rate (ORR) (partial response [PR] or better)

• To determine duration of response (DOR)

• To determine time to progression (TTD)

- To determine safety
- To determine overall survival (OS)

## 4.3 **Additional Objectives**

Not applicable

## 4.4 **Study Design**

only and subject to the ic This is a phase 2, open-label, single arm, multicenter study to evaluate the efficacy and safety of ixazomib plus lenalidomide and dexamethasone in Japanese patients with relapsed and/or refractory multiple myeloma (MM). The patient population will consist of adult men and women who have a confirmed diagnosis of MM, who have received 1 to 3 prior lines of therapy, and who meet other outlined eligibility criteria (see Section 7.0). Approximately 30 patients will be enrolled in the study.

General eligibility criteria may be assessed prior to the formal Screening period if it is part of standard clinical practice. However, per the Schedule of Events, formal screening will occur during the Screening period, which may last for up to 28 days prior to enrollment. A Takeda clinician will confirm patient eligibility prior to enrollment. Determination of disease progression as an entry criterion may be based on patient data obtained during or following the patient's most recent prior antineoplastic therapy.

Patients will receive study drug (ixazomib 4.0 mg) on Days 1, 8, and 15 plus lenalidomide (25 mg) on Days 1 through 21 and dexamethasone (40 mg) on Days 1, 8, 15, and 22 of a 28day cycle. Patients may continue to receive treatment until progressive disease (PD) or unacceptable toxicity, whichever comes first. Dose modifications may be made based on toxicities. Patients with a low creatinine clearance < 60 mL/min will receive a reduced lenalidomide dose of 10 mg. The lenalidomide dose may be escalated to 15 mg after 2 cycles if the patient is not responding to treatment and is tolerating the treatment. If renal function normalizes (ie, creatinine clearance ≥ 60 mL/min) and the patient continues to tolerate this treatment, lenalidomide may then be escalated to 25 mg.

Patients will be seen at regular treatment cycle intervals while they are participating in the study: four times a treatment cycle for the first 2 cycles, twice a treatment cycle for the 3rd

150 NSE

cycle, and then once a treatment cycle for the remainder of their participation in the active treatment and, if applicable, the PFS (every 4 weeks) and OS (every 12 weeks) follow-up phases of the study.

Response will be assessed by investigator according to the IMWG criteria for all patients every 4 weeks until PD. Central laboratory data will be used for serum M-protein, urine M-protein and serum free light chain. All patients will be followed for survival after progression. Patients will be contacted every 12 weeks until death or termination of the study by the sponsor.

Patients will attend an End of Treatment (EOT) visit approximately 30 days after receiving their last dose of study treatment (ixazomib, lenalidomide or dexamethasone) and will continue to be followed for other follow-up assessments specified in the Schedule of Events. Patients discontinuing study treatment prior to PD will continue to be assessed for PD during the PFS follow-up portion of the study.

Analysis is planned to be performed twice during the study. The primary analysis is planned to be performed using the data obtained at approximately 12 months from the enrollment of the last patient. The final analysis is planned to be performed after the final database lock en ational at a seed a for non-commercial use only all a property of Takeda. For non-commercial use only a seed a for non-commercial use only a seed a se using the data obtained at approximately 24 months from the enrollment of the last patient. The timing of analysis may be changed or additional analysis may be added upon request of

# 5.0 ANALYSIS ENDPOINTS

# Primary Efficacy Endpoint

VGPR or better rate in response-evaluable analysis set

# Secondary Efficacy Endpoints

- PFS, defined as the time from the date of first study drug administration to the date of first documentation of PD or death from any cause, whichever occurs first
- ORR
- DOR, defined as the time from the date of first documentation of response to the date of first documentation of PD
- TTP, defined as the time from the date of first study drug administration to the date of first documentation of PD
- Safety including treatment-emergent adverse events (TEAEs), laboratory parameters, and vital signs
- OS, defined as the time from the date of first study drug administration to the date of death

# 6.0 DETERMINATION OF SAMPLE SIZE

Assuming the expected VGPR or better rate is 48.1% and the threshold rate is 39.0% based on the results of Study C16010, a sample size of 27 would be necessary to provide a point estimate of VGPR or better rate higher than the threshold rate with 80% probability. Assuming a drop-out ratio of 10%, the target number of patients has been set to 30. The expected response rate and the threshold assumptions are based on VGPR or better rate in ixazomib + LenDex arm and placebo + LenDex arm in Study C16010 (intent-to-treat population, primary analysis).

# 7.0 METHODS OF ANALYSIS AND PRESENTATION

# 7.1 General Principles

# 7.1.1 Study Definitions

The following definitions and calculation formulas will be used.

- Descriptive statistics: Number of subjects, mean, standard deviation, maximum, minimum, and quartiles
- Frequency distributions: Number of subjects and percentage (of nonmissing) percategory
- Baseline body surface area (m<sup>2</sup>): square root of (baseline height \* baseline weight / 3600)
- Time since initial diagnosis to first dose at study entry (months): (first dose date date of initial diagnosis + 1) / (365.25 / 12)
- Relapsed patients: Patients who relapsed from at least 1 previous treatment but were not refractory to any previous treatment. Patients who progress after 60 days from the last dose of a given therapy will be considered relapsed.
- Refractory patients: Patients who were refractory to at least 1 previous treatment but were not relapsed to any previous treatment. Refractory disease is defined as disease progression on treatment or progression within 60 days after the last dose of a given therapy.
- Refractory and relapsed patients: Patients who were relapsed from at least 1 previous treatment and additionally were refractory to at least 1 previous treatment.
- Primary refractory patients: Patients who are refractory to all lines of previous therapy (i.e., best response to prior therapy is SD or disease progression on all lines of therapy).
- Time since last transplant to first dose at study entry (months): (first dose date start date of prior transplant) / (30.4375)
- Relative dose intensity: 100 \* (total amount of dose taken) / (total prescribed dose of treated cycles), where total prescribed dose equals [dose prescribed at enrollment \* number of prescribed doses per cycle \* the number of treated cycles]
- Extent of Exposure (cycles) is based on the number of treated cycles.
- Extent of Exposure (days): date of last dose date of first dose + 1
- Percent drug compliance (%): (study drug taken in mg) / (study drug expected to be taken in mg) \*100%
- Treatment-emergent adverse event (TEAE): Any adverse event that occurs after administration of the first dose of any study drug through 30 days after the last dose of any study drug
- If corrected calcium is not reported directly, it can be calculated using the following formula:
  - ➤ Corrected Calcium (mmol/L): serum calcium (mmol/L) + 0.0200 \* (40 serum albumin (g/L))

# **Definition of Study Visit Windows**

Plicable Leiths of Use Unless otherwise specified, the baseline value is defined as the value collected at the time closest to, but before, the start of study drug administration.

All data will be categorized on the basis of the scheduled visit at which they are collected.

# 7.1.3 Significance Level and Confidence Coefficient

Confidence coefficient: 95% (two-sided)

## 7.2 **Analysis Sets**

In this study, the following three analysis sets are defined.

- FAS: All subjects who received at least one dose of the study drug during the treatment period. Subjects will be excluded from FAS if the following criterion is met:
  - No study drug received
- Response-evaluable analysis set: All FAS subjects with measurable disease at baseline, and at least one post baseline response assessment. Measurable disease is defined by at least 1 of the following 3 measurements based on central laboratory data: serum Mprotein  $\geq 1$  g/dL ( $\geq 10$  g/L), urine M-protein  $\geq 200$  mg/24 hours, and serum free light chain assay where involved free light chain level  $\geq 10 \text{ mg/dL}$  ( $\geq 100 \text{ mg/L}$ ), provided that the serum free light chain ratio is abnormal.

Subjects will be excluded from the response-evaluable analysis set if any of the following criteria are met:

- No measurable disease at baseline
- No post-baseline assessment
- No study drug received
- Safety analysis set: All subjects who received at least one dose of the study drug during the treatment period. Subjects will be excluded from the safety analysis set if the following criterion is met:
- Property of Lakeda No study drug received

# 7.3 Disposition of Subjects

# 7.3.1 Study Information

Analysis Set: All Subjects Who Signed the Informed Consent Form

Analysis

Variable(s): Date First Subject Signed Informed Consent Form

Date of Last Subject's Last Visit/Contact

MedDRA Version
WHO Drug Version

SAS Version Used for Creating the Datasets

Analytical

Method(s): (1) Study Information

Study information shown in the analysis variables section will be provided.

# 7.3.2 Number of Subjects Who Entered the Treatment Period by Site

Analysis Set: All Subjects Who Entered the Treatment Period

Analysis

Variable(s): Status of Entrance into the Treatment [Entered]

Period

Stratum: Site [Site numbers will be used as

categories]

Analytical

Method(s): (1) Number of Subjects Who Entered the Treatment Period by Site

Frequency distribution will be provided for each stratum.

# 7.3.3 Disposition of Subjects

Analysis Set: All Subjects Who Entered the Treatment Period

Analysis

Variable(s): Study Drug Completion Status [Ongoing on Treatment, Prematurely

Discontinued Study Drug]

Reason for Discontinuation of [Adverse Event, Lost to Follow-up,

Study Drug Progressive Disease, Protocol

Violation, Study Terminated by Sponsor, Withdrawal by Subject,

Other]

Subjects that have Participated in OS

Follow-up

Subjects that have Participated in [Yes, No]

PFS Follow-up

Completion Status of the Follow-up [Completed Follow-up Period,

Period Prematurely Discontinued Follow-up

Period]

[Lost to Follow-up, Study Terminated

Reason for Discontinuation of the

Follow-up Period by Sponsor, Withdrawal by Subject,

Other]

Analytical

Method(s): (1) Disposition of Subjects

Frequency distributions will be provided.

# 7.3.4 Protocol Deviations and Analysis Sets

# 7.3.4.1 Protocol Deviations

Analysis Set: All Subjects Who Entered the Treatment Period

**Analysis** 

Variable(s): Significant Protocol [Entry Criteria, Concomitant Medication,

Deviation Procedure Not Performed Per Protocol, Study

Medication, Withdrawal Criteria, Good Clinical

Practice]

Analytical

Method(s): (1) Protocol Deviations

Frequency distribution will be provided for each deviation category. A subject who has several deviations will be counted once in each appropriate category. A subject who has several deviations that can be classified into the

same category will be counted only once.

# 7.3.4.2 Analysis Sets

Analysis Set: All Subjects Who Entered the Treatment Period

Analysis

Variable(s): Handling of Subjects [Categories are based on the

specifications in Section 7.2

Analytical

Method(s):

[Included]

[Inclu

# Race property of Lakedai. **Demographic and Other Baseline Characteristics**

# 7.4.1.1 Demographic and Other Baseline Characteristics

 $Min \le - \le 65, 65 < - \le 75,$ 

75 < - <= Max

[Male, Female]

[Hispanic or Latino, Not Hispanic or

Latino, Not Reported]

[White, Black or African American,

Native Hawaiian or Other Pacific

Islander, Asian (Asian Indian), Asian

(Chinese), Asian (Japanese), Asian (Korean), Asian (Other), Asian (Not

Reported), American Indian or

Alaska Native, Not Reported, Other]

Dose at Study Entry (months)

ISS Stage at Initial Diagnosis [I, II, III, Unknown]

**Patient Population Categories** [Relapsed Patients,

Refractory Patients,

le Leithe Of Use Refractory and Relapsed Patients]

Type of Myeloma at Initial Diagnosis

**IgG** [Kappa, Lambda, Biclonal,

Unknown]

[Kappa, Lambda, Biclonal, ] **IgA** 

Unknown]

[Kappa, Lambda, Biclonal, IgD

Unknown]

IgE [Kappa, Lambda, Biclonal,

Unknown \

[Kappa, Lambda, Biclonal, **IgM** 

Unknown]

**Biclonal** Kappa, Lambda, Biclonal,

Unknown]

[Kappa, Lambda, Biclonal, Unknown

Unknown]

Other [Kappa, Lambda, Biclonal,

Unknown]

Durie-Salmon Stage at Initial [IA, IB, IIA, IIB, IIIA, IIIB,

Diagnosis Unknown] Lines of Prior Therapy [1, 2, 3]

Evidence of Lytic Bone Disease at [Yes, No, Unknown]

**Initial Diagnosis** 

Evidence of Extramedullary Disease [Yes, No, Unknown]

at Initial Diagnosis


Patients with a Bone Marrow

Transplant or Stem Cell Transplant

Type of Transplant Procedure [Allogenic, Autologous, Both,

Unknown]

Time Since Last Transplant to First

Dose at Study Entry (months)

Type of Prior Regimens [Velcade Contained,

Thalidomide Contained,

Thalidomide Refractory,

Lenalidomide Contained,

icable Terms of Use Corticosteroids Contained.

Dexamethasone,

Prednisone.

Other,

Carfilzomib Contained,

Melphalan Contained,

Other]

Type of Last Prior Regimen

[Velcade Contained,

Thalidomide Contained,

Thalidomide Refractory,

Lenalidomide Contained,

Corticosteroids Contained,

Dexamethasone,

Prednisone,

Other.

Carfilzomib Contained,

Melphalan Contained,

Other]

Patient was Relapsed on Last Prior

Therapy

Patient was Refractory on Last Prior

[Yes, No]

[Yes, No]

Therapy

Time Since Last Dose of Prior

Therapy to First Dose at Study Entry

(months)


Best Response to Prior Therapy

[Complete Response, Partial

Response, Stable Disease,

Progressive Disease, Unable to

Assess, Unknown]

Time Since Disease Progression on

Prior Therapy to First Dose at Study

Entry (months)

Patients with Prior Radiation

Time Since Last Prior Radiation to

First Dose at Study Entry (months)

Patients with Prior Surgery or Non-

**Radiation Procedures** 

Time Since Last Prior Surgery or Non-Radiation Procedure to First

Dose at Study Entry (months)

Prior IMiD Therapy [Exposed,

> Thalidomide, Lenalidomide, Pomalidomide.

Naive]

[Yes, No]

Patient was Refractory to Any Prior

IMiD Therapy

Prior Proteasome Inhibitor Therapy [Exposed

Velcade,

Carfilzomib,

Naive]

Patient was Refractory to Any Prior [Yes, No]

Proteasome Inhibitor Therapy

**Primary Refractory Patients** 

[Progression Disease, Stable Disease]

ISS Stage for Myeloma at Study [I, II, III]

Entry

Evidence of Lytic Bone Disease [Present, Absent, Unknown]

Extramedullary Disease at Study

Entry

Serum M-Protein (g/L)

Urine M-Protein (g/24h)

Serum Creatinine (mg/dL)  $[Min \le - \le 2, 2 \le - \le Max]$ 

Serum Albumin (g/L)  $[Min \le - <35, 35 \le - <=Max]$ 

 $\beta_2$ -microglobulin (mg/L)  $[Min \le - <3.5, 3.5 \le - <5.5,$ 

 $5.5 \le - \le Max$ 

[Yes, No, Unknown]

Creatinine Clearance (mL/min)  $[Min \le - <30, 30 \le - <60,$ 

 $60 \le -490, 90 \le -4 \le Max$ 

Corrected Calcium (mmol/L)

Baseline ECOG Performance Status

[0, 1, 2, 3, 4]

Baseline Hemoglobin (g/L)

Analytical


Method(s): (1) Summary of Demographics and Baseline Characteristics

icable reins of Use applicable applicable applicable to the applic Frequency distributions for categorical variables and descriptive statistics for

continuous variables will be provided.

7.4.1.2 Baseline Bone Marrow Evaluation and Extramedullary Disease Assessment

Full Analysis Set Analysis Set:

Analysis


Variable(s): Bone Marrow Aspiration

Number of Patients with Bone

Marrow Aspiration

Number of Patients with Adequate

Sample for Interpretation

% Plasma Cells [Available, Unable to Detect,

Not Available]

Bone Marrow Biopsy

Number of Patients with Bone

Marrow Biopsy

Number of Patients with Adequate

Sample for Interpretation

% Plasma Cells [Available, Unable to Detect,

Not Available]

% Marrow Cellularity [Available, Not Available]

Marrow Cellularity Status [Hypocellular, Hypercellular,

Normocellular, Unable to Assess]

Ommunohistochemistry or

Immunofluorescence for

Kappa/Lambda Ratio Performed

[Yes, No, Not Applicable]

Ratio Determined by Analysis of a

Minimum of 100 Plasma Cells

[Yes, No, Not Applicable]

% Plasma Cells in Bone Marrow

Kappa/Lambda Ratio

Bone Marrow Cytogenetic Results

Sample Collected? [Yes, No, Not Applicable]

Method of Assessment [Conventional/Karotype,

Molecular/FISH, Both]

Cytogenetic Results

(Conventional/Karotype) [Normal, Abnormal, Indeterminate]

Cytogenetic Results

e Terms of Use (Molecular/FISH) [Normal, Abnormal, Indeterminate]

Abnormality of Chromosomal

Aberrations

Subjects with Any Chromosomal [Del 13 or -13q, Del 17 or -17p]

Abnormalities t(4;14), t(6;14), t(8;14), t(11;14),

t(12;14), t(14;16), t(14;20),

Hyperdiploidy, Hypodiploidy,

Non-hyperdiploidy,

1q amplification, 1q deletion, Other]

Cytogenetic Results [High Risk, Standard, Not Available]

Skeletal Survey

Result Within Normal Limits, Abnormal]

Lytic Bone Lesions Present [Yes, No, Indeterminate]

Imaging (Computed Tomography)

Result [Within Normal Limits, Abnormal]

Plasmacytomas Present [Yes, No, Indeterminate]

Imaging (Magnetic Resonance

Imaging)

Result [Within Normal Limits, Abnormal]

Plasmacytomas Present [Yes, No, Indeterminate]

Imaging (Positron Emission

Tomography)

PET Activity [FDG Positive, FDG Negative,

Indeterminate]

Property of Takeda. Fo Subjects with Plasmacytomas [Liver (Visceral), Lung (Visceral),

Node, Soft Tissue, Lytic Bone,

Other]

Number of Plasmacytomas

[1, 2, >=3]

Soft Tissue Plasmacytomas Total

Size (cm<sup>2</sup>)

Lytic Bone Plasmacytomas Total

Size (cm<sup>2</sup>)

Analytical

Method(s): (1) Baseline Bone Marrow Evaluation and Extramedullary Disease Assessment

to the applicable Terms of Use 5, r Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided.

7.4.1.3 Disease Specific History – IMiD and Proteasome Inhibitor

Analysis Set: Full Analysis Set

Analysis

Variable(s): Exposed to Prior IMiD Therapy

Lenalidomide

Lenalidomide Refractory

Best Response [CR, PR, SD, PD, Unable to Assess,

Unknown]

Thalidomide

Thalidomide Refractory

Best Response [CR, PR, SD, PD, Unable to Assess,

Unknown]

Pomalidomide

Pomalidomide Refractory

Best Response [CR, PR, SD, PD, Unable to Assess,

Unknown]

Exposed to Prior Proteasome

Inhibitor Therapy

Velcade Refractory

Best Response [CR, PR, SD, PD, Unable to Assess,

Unknown]

Carfilzomib

Carfilzomib Refractory

Best Response [CR, PR, SD, PD, Unable to Assess,

Unknown]

(1) Disease Specific History – IMiD and Proteasome Inhibitor

Frequency distributions for categorical variables will be provided. For the analysis variables "Exposed to Prior IMiD Therapy", "Lenalidomide",
"Thalidomide", "Pomalidomide", "Exposed to Prior Proteasome Inhibitor Therapy", "Velcade", and "Carfilzomib", the denominators for the percentages will be the number of subjects in FAS. For the analysis variables "Lenalidomide Refractory", "Thalidomide Refractory", "Pomalidomide Refractory", "Velcade Refractory", and "Carfilzomib Refractory", the denominators for the percentages will be the number of subjects who were exposed to the specified therapy (Lenalidomide, Thalidomide, Pomalidomide, Velcade, or Carfilzomib). For the analysis variable "Best Response", the denominators for the percentages will be the number of subjects who were refractory to the specified therapy (Lenalidomide, Thalidomide, Pomalidomide, Velcade, or Carfilzomib).

7.4.1.4 Summary of Baseline Measurable Status in Subjects with only Abnormal Baseline Free Light Chain

Analysis Set: Full Analysis Set

Analysis

Variable(s): Free Light Chains (no Heavy Chain)

Measureable

Measureable by FLC only

Non-measureable

Analytical

Method(s): (1) Summary of Baseline Measurable Status in Subjects with only Abnormal

Baseline Free Light Chain

Frequency distributions for categorical variables will be provided.

7.4.1.5 Summary of New Primary Malignancy

Analysis Set: Full Analysis Set

**Analysis** 

Variable(s): Subjects with any New Primary

Malignancy

New Primary Malignancy Disease

Type (On Treatment) [Categories will be based on actual

data]

New Primary Malignancy Disease

Type (Follow-up) [Myelodysplastic syndrome,

insofuse Acute myeloid leukaemia or related precursor neoplasm, Precursor lymphoid neoplasm, Mature B-cell neoplasm, Mature T-cell and NK-cell neoplasm. Hodgkin lymphoma, Solid Tumor, Otherl

Analytical

Method(s):

(1) Summary of New Primary Malignancy

Frequency distributions will be provided. Summaries will be provided using the new primary malignancy disease type and its detailed categories, where the detailed categories will be sorted alphabetically.

#### 7.5 **Medical History and Concurrent Medical Conditions**

Safety Analysis Set Analysis Set:

**Analysis** 

Variable(s): Medical History

**Concurrent Medical Conditions** 

Analytical

Property of Takeda

(1) Medical History by Verbatim Term Method(s):

> (2) Concurrent Medical Conditions by System Organ Class and Preferred Term

Frequency distributions will be provided.

For (1), summary will be provided using verbatim terms. A subject with multiple occurrences of medical history within a verbatim term will be counted only once in that verbatim term.

For (2), MedDRA dictionary will be used for coding. Summary will be provided using SOC and PT, where SOC and PT will be sorted in decreasing frequency. A subject with multiple occurrences of concurrent medical condition within a SOC will be counted only once in that SOC. A subject with multiple occurrences of concurrent medical condition within a PT will

be counted only once in that PT.

#### 7.6 **Medication History and Concomitant Medications**

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Concomitant Medications

Analytical

(1) Concomitant Medications by ATC Pharmacological Subgroup and WHO Method(s):

Generic Term

Frequency distributions will be provided. Concomitant medications are defined as medications with start dates occurring on or after date of first dose and before date of last dose + 30 days. WHO Drug dictionary will be used for coding. Summaries will be provided using ATC pharmacological subgroup and WHO generic term. ATC pharmacological subgroup will be sorted alphabetically and WHO generic term will be sorted in decreasing frequency based on the number of reports. A subject who has been administered several medications with the same WHO generic term will be counted only once for that WHO generic term.

#### Study Drug Exposure and Compliance 7.7

7.7.1.1 Study Drug Exposure and Compliance

Analysis Set: Safety Analysis Set

Analysis

Total Amount of Doses Taken (mg) Variable(s):

Total Number of Doses Taken

Number of Treated Cycles [>=1, >=2, >=3, >=4, >=5, >=6, >=7,

>=8, >=9, >=10, >=11, >=12, >=13,

>=14, >=15, >=16, >=17, >=18,

>=19, >=20, >=21, >=22, >=23,

>=241

Property of Takedai. Fr [Min<= - <50, 50<= - <80, Relative Dose Intensity (%)

 $80 \le -100, 100, 100 \le -100$ 

Extent of Exposure (cycles) [1<= - <=3, 4<= - <=6, 7<= -<=9,

10<= - <=12, 13<= - <=15,

16<= - <= 18, 19<= - <= 21,

22<= - <=24, 24< - <=Max]

Extent of Exposure (days)

he Leims of Use

$$100 < - <= Max$$

Analytical

Method(s): (1) Study Drug Exposure and Compliance – Ixazomib

(2) Study Drug Exposure and Compliance – Lenalidomide

(3) Study Drug Exposure and Compliance – Dexamethasone

(4) Study Drug Exposure and Compliance – Combination (Ixazomib Lenalidomide, Dexamethasone)

Frequency distributions for categorical variables and descriptive statistics for continuous variables will be provided. For (4), only the number of treated cycles, extent of exposure (cycles), and extent of exposure (days) will be provided.

Mean and 95% CI plots of changes over time will be provided for the relative dose intensity. A treated cycle is defined as a cycle in which the patients received any amount of Ixazomib for (1), Lenalidomide for (2),

Dexamethasone for (3), and any of Ixazomib, Lenalidomide, Dexamethasone for (4).

## 7.7.1.2 Dose Modifications

Safety Analysis Set Analysis Set:

Analysis

Dose Modification

[No Action Taken, Reduced

Prescribed, Reduced Non-Prescribed, Increased Prescribed, Increased non-Prescribed, Held, Missed, Delayed,

Discontinued Permanently]

Cycle Delayed Action on Drug Number of Subjects with at least 1 Dose Reduction Number of Subjects with at least 2 Dose Reduction

(1) Dose Modifications – Ixazomib

(2) Dose Modifications – Lenalidomide

(3) Dose Modifications – Dexamethasone

insofuse Frequency distributions will be provided for overall, for every cycle from Cycle 1 to 18, and for Cycles 1-6, 7-12, 13-18, 19-21, 22-24, >=25. The analysis variable "dose modification" includes reduced prescribed, reduced non-prescribed, increased prescribed, increased non-prescribed, delayed, and discontinued permanently. For the analysis variable "Action on Drug", a 📈 🔾 subject will be counted once for each unique reason for dose modification that they have had over the course of the study. For "Action on Drug", the numerators for the percentages are the number of subjects with a dosing Abe as a present of takeda. For noncommercial use only and subject to modification and the denominators are the total number of subjects with nonmissing dosing data. Dose reduction is defined as a prescribed reduction in

#### **7.8 Efficacy Analysis**

#### 7.8.1 **Primary Efficacy Endpoint(s)**

#### 7.8.1.1 Primary Analysis

Analysis Set:

Analysis

Variable(s):

Analytical

Method(s):

VGPR
Overall Response (CR+PR (including sCR and VGPR))
VGPR or better (CR+VGPR)
SD
'D

1e VGPR or better (ervals w''' intervals will be provided in the response-evaluable analysis set as the primary analysis. The response rate and the 2-sided 95% confidence intervals will be provided for each analysis variable based on the confirmed best response.

The response rates and the 2-sided 95% confidence intervals will also be summarized based on the unconfirmed best response and the best response (confirmed or unconfirmed) at the end of each cycle (from Cycle 1 to Cycle 24).

The ORR is defined as the proportion of patients who achieved PR or better. Stacked bar graph will be provided for ORR (confirmed or unconfirmed) and ORR (confirmed) at the end of each cycle and overall.

#### Sensitivity Analysis

Full Analysis Set

Analysis

Variable(s): CR

**sCR** 

PR

**VGPR** 

Kerms of Use

Overall Response (CR+PR (including sCR and VGPR))

VGPR or better (CR + VGPR)

SD

PD

Not Evaluable

Analytical

Method(s):

To check the robustness of the results, the same analyses as those in Section 7.8.1.1 will be performed using FAS, except for the summary based on the best response (confirmed or unconfirmed) at the end of each cycle and the stacked bar graphs for ORR. Non-evaluable subjects in FAS will only be included in the denominator when calculating the response rates. The VGPR or better (CR + VGPR) rate and the 2-sided 95% confidence intervals will be provided in FAS as the sensitivity analysis for the primary analysis. Non-evaluable subjects in FAS will be included in the analysis as Use only and not VGPR or CR.

## **Secondary Efficacy Endpoint(s)**

#### 7.8.2.1 Progression-free Survival

Full Analysis Set Analysis Set:

**Analysis** 

Variable(s):

Analytical

Method(s):


For the PFS, the Kaplan-Meier curve [and the 25th, 50th (median), and 75th percentiles, if estimable] will be calculated with their 2-sided 95% CIs in FAS. Kaplan-Meier estimates will also be calculated at 6 months, 9 months, 12 months, 18 months, and 24 months with their 2-sided 95% CIs. The median follow-up time in months and its 2-sided 95% CI will also be provided.

PFS is defined as the time from the date of first study drug administration to the date of first documentation of PD or death from any cause, whichever occurs first. The number of subjects with events and the number of subjects censored will be provided as well as the reason for censoring. Patients without documentation of PD will be censored at the date of the last response assessment that is SD or better. The details regarding the handling of missing assessments and censoring are presented in the table below.

| Situation | Date of Progression | Outcome |
|--------------------------------------|-------------------------|------------|
| Situation | G | Outcome |
| | or Censoring | |
| No baseline and/or no post baseline | Date of first dose | Censored |
| assessment, no subsequent | | 16 |
| anticancer therapy after study | | 2/6 |
| treatment, no death | | ··COL |
| Disease progression documented | Date of next | Progressed |
| between scheduled visits | scheduled visit | |
| No documented death or disease | Date of last adequate | Censored |
| progression | assessment <sup>1</sup> | |
| Lost to follow-up, withdraw | Date of last adequate | Censored |
| consent before any documented | assessment <sup>1</sup> | |
| death or disease progression | 250 | |
| Death or progression after more | Date of last adequate | Censored |
| than 1 missed visit <sup>2</sup> | assessment <sup>1</sup> | |
| Alternate antineoplastic therapy | Date of last adequate | Censored |
| started prior to disease progression | assessment prior to | |
| | starting alternate | |
| o (C)lo | antineoplastic therapy | |
| Death before first post baseline | Date of death | Progressed |
| assessment | | |
| Death between adequate assessment | Date of death | Progressed |
| visits | | |

Adequate disease assessment is defined as there is sufficient data to evaluate a subject's disease status.

<sup>2</sup>: Death or progression occurs more than 90 days from previous adequate assessment.

## 7.8.2.2 Duration of Response

Analysis Set: Responders in the Full Analysis Set

Analysis

Variable(s): DOR

Analytical

Method(s): For the DOR, the Kaplan-Meier curve [and the 25<sup>th</sup>, 50<sup>th</sup> (median), and 75<sup>th</sup>

percentiles, if estimable will be calculated with their 2-sided 95% CIs for the

DOR is defined as the time from the date of first documentation of response to the first documentation of PD. Responders without documentation of PD. Will be censored at the date of their last response better. The number of a 1. censored will be provided as well as the reason for censoring. For the analysis of DOR, "response" will be defined as (1) VGPR or better Use only and subject (2) ORR (3) CR and the same analysis will be performed for each type of response.

#### 7.8.2.3 Time to Progression

Full Analysis Set Analysis Set:

**Analysis** 

Variable(s): TTP

Analytical

Method(s):

Proberty of Lakeda.

For the TTP, the Kaplan-Meier curve [and the 25th, 50th (median), and 75th percentiles, if estimable] will be calculated with their 2-sided 95% CIs in FAS. Kaplan-Meier estimates will also be calculated at 6 months, 9 months, 12 months, 18 months, and 24 months with their 2-sided 95% CIs. TTP is defined as the time from the date of first study drug administration to the date of first documentation of PD. Patients without documentation of PD at the time of analysis will be censored at the date of their last response assessment that is SD or better. Patients with no response assessment will be censored at the first day of administration. Patients who do not experience progression and start new systemic therapy for multiple myeloma will be censored at the date of their last response assessment that is SD or better. The number of subjects with events and the number of subjects censored will be provided as well as the reason for censoring.

#### 7.8.2.4 Overall Survival

Analysis Set: Full Analysis Set

Analysis

Variable(s): OS

Analytical

For the OS, the Kaplan-Meier curve [and the 25th, 50th (median), and 75th Method(s):

> percentiles, if estimable] will be calculated with their 2-sided 95% CIs in FAS. Kaplan-Meier estimates will also be calculated at 6 months, 9 months, 12 months, 18 months, and 24 months with their 2-sided 95% CIs. The median follow-up time in months and its 2-sided 95% CI will also be

provided.

OS is defined as the time from the date of first study drug administration to the date of death. Subjects without documentation of death at the time of the analysis will be censored at the date when they were last known to be alive. The number of deaths and the number censored will be provided as well as

the reason for censoring.

# Additional Efficacy Endpoint(s)

#### 7.8.3.1 Best M-Protein Response to Treatment

Response-evaluable Analysis Set Analysis Set:

Analysis

Best M-Protein Response Variable(s):

Property of Lakedai. For Response Category [100% Reduction, Categories:

Immunofixation Negative,

>=90% Reduction,

>=50% Reduction]

[90 - <100% Reduction,

75 - <90% Reduction.

50 - <75% Reduction,

25 - <50% Reduction]

[<25% Reduction to <25% Increase,

>=25% Increase]

No Post-Baseline Assessment of Measurable M-Protein

Analytical

Method(s):

Frequency distribution will be provided. For subjects with measurable serum M-protein at baseline, the best M-protein response is the percent change from baseline to best (lowest) value post-baseline in serum M-protein. For subjects with non-measurable serum M-protein, but measurable urine M-protein, the best M-protein response is the percent change from baseline to best (lowest)? value post-baseline in urine M-protein. Mean and standard deviation plots of changes over time will be provided for observed values and percent changes from baseline. A waterfall plot will be provided for the percent changes from TO THE DE baseline.

Page 31 of 46

#### 7.8.3.2 Time to Response

Responders in the Response-evaluable Analysis Se Analysis Set:

Full Analysis Set

Analysis

VGPR or better (CR + VGPR) Variable(s):

Overall Response

Analytical

For the time to response, the Kaplan-Meier curve [and the 25<sup>th</sup>, 50<sup>th</sup> (median), Method(s):

> and 75th percentiles, if estimable will be calculated with their 2-sided 95% CIs. Kaplan-Meier estimates will also be calculated at 6 months, 9 months,

12 months, 18 months, and 24 months with their 2-sided 95% CIs.

Time to response is defined as the time from the date of first study drug administration to the date of first documentation of the confirmed response indicated in the analysis variable. Responders are defined as subjects with documentation of a confirmed response of the analysis variable. The number of subjects with events and the number of subjects censored will be provided as well as the reason for censoring.

The same analyses will be performed using FAS.

## 7.8.3.3 Duration of Follow-up

Analysis Set: Full Analysis Set

**Analysis** 

Variable(s): Duration of Follow-up

Analytical

For the duration of follow-up, the Kaplan-Meier curve [and the 25<sup>th</sup>, 50<sup>th</sup> Method(s):

(median), and 75<sup>th</sup> percentiles, if estimable] will be calculated with their 2-sided 95% CIs. Kaplan-Meier estimates will also be calculated at 6 months, 9 months, 12 months, 18 months, and 24 months with their 2-sided 95% CIs. The median follow-up time in months and its 2-sided 95% CI will also be provided.

Duration of follow-up is defined as time from the date of first study drug administration to the date of death or last known visit. The number of subjects with events and the number of subjects censored will be provided as well as the reason for censoring.

#### 7.8.4 Statistical/Analytical Issues

7.8.4.1 Adjustments for Covariates

Not applicable.

7.8.4.2 Handling of Dropouts or Missing Data

Censoring rules have been described in each applicable section.

7.8.4.3 Multicenter Studies

Treatment-by-center interaction will not be explored since this study is a single-arm study.

7.8.4.4 Multiple Comparison/Multiplicity

Not applicable.

7.8.4.5 Use of an "Efficacy Subset" of Subjects

In addition to analyses on the primary endpoint using the response-evaluable analysis set, a secondary analysis will also be performed using the FAS to examine the robustness of the results.

7.8.4.6 Active-Control Studies Intended to Show Equivalence or Non-Inferiority Not applicable.

7.8.4.7 Examination of Subgroups

Analysis Set: Response-evaluable Analysis Set

Full Analysis Set

Analysis

Variable(s): CR

sCR

PR

**VGPR** 

Overall Response (CR+PR (including sCR and VGPR))

VGPR or better (CR + VGPR)

SD

PD

Subgroup(s): Age (years)  $[Min \le - \le 65, 65 \le -$ 

75 < - <= Max

Sex [Male, Female]

Cytogenetic Risk [High Risk {(del17); t(4;14);

t(14;16)}, Non-High Risk]

ISS Stage for Myeloma at Study [I, II, III]

Entry

Lines of Prior Therapy [1, 2 or 3]

Prior Proteasome Inhibitor Therapy [Exposed, Naive]

Prior IMiD Therapy [Exposed, Naive]

Thalidomide Refractory [Yes, No]
Refractory to Any Line of Prior [Yes, No]

Therapy

Patient was Refractory on Last Prior [Yes, No]

Therapy

Relapsed and/or Refractory [Relapsed, Refractory, Relapsed and

Refractory]

Prior Veloade Therapy [Exposed, Naive]

Creatinine Clearance (mL/min)

 $[Min \le - <60, 60 \le - <=Max]$ 

 $[Min \le - <50, 50 \le - <=Max]$ 

Baseline ECOG Performance Status [0 or 1, 2]

Prior Lenalidomide Therapy [Exposed, Naive]
Prior Thalidomide Therapy [Exposed, Naive]

Analytical

Method(s): The same analyses as those in Sections 7.8.1.1 and 7.8.1.2 will be performed

with the confirmed best response for each subgroup. A forest plot will be produced using the VGPR or better (CR+VGPR) rate and the 2-sided 95%

confidence intervals.

#### 7.8.4.8 Examination of Subgroups – Summary Table

Analysis Set: Response-evaluable Analysis Set

Full Analysis Set

Analysis

Variable(s): ORR

> VGPR or better CR or better

Subgroup(s): Age (years)

Sex

Cytogenetic Risk

[Min<= - <=65, 65< - <=75, 75< - <=Max] Male, Female] Not Availah igh F High Risk, High Risk (del17), High Risk t(4;14), High Risk t(14;16)]

[0, 1, 2]Baseline ECOG Performance Status

Prior Lines of Therapy per Takeda

review with SCT, without SCT,

with SCT, without SCT,

3,

with SCT, without SCT]

Relapsed/Refractory Type [Relapsed, Refractory,

Relapsed and Refractory,

Primary Refractory]

Prior Proteasome Inhibitor [Exposed, Naive,

Refractory,

Vc-Refractory (Takeda),

CFZ-Refractory (Takeda)]

Prior IMiD [Exposed, Naive,

Refractory,

Thal-Refractory (Takeda), Len-Refractory (Takeda)]

ISS stage at Study Entry [I, II, III]

Best Response [>=CR, >=VGPR, >=PR, SD, PD]

Creatinine Clearance (mL/min)  $[Min \le - <50, 50 \le - <=Max]$ 

 $Min \le - <50, 50 \le - <60,$ 

 $60 \le - \le Max$ 

**CONFIDENTIAL** 

Property of Takedai. For

[Min<= - <60, 60<= - <=Max]

1 Prior Line with SCT

High Risk

ISS 3

Prior IMiD [Exposed, Naive]
Thalidomide [Exposed, Naive]
Lenalidomide [Exposed, Naive]

Maintenance Therapy [Yes, No]

Time from SCT to First Dose  $[0 \le -12, 12 \le -24, 24 \le -36,$ 

(Months) 36<= - <= Max]
Prior PI [Exposed, Naive]

1 Prior Line with SCT

Single vs. Double SCT [Single SCT, Double SCT]

With Velcade + Thalidomide [Yes, No]
With Velcade + Lenalidomide [Yes, No]

Best Response on Prior SCT [CR, PR, SD or PD]

ECOG [0, 1]

Low Bone Marrow Cellularity [Yes, No, Missing]

Cytogenetic Risk [Not Available,

1 Line with SCT, Others]

Analytical

Method(s): Frequency distributions for each analysis variable will be provided for each

subgroup.

#### 7.9 Pharmacokinetic/Pharmacodynamic Analysis

## 7.9.1 Pharmacokinetic Analysis

Not applicable.

## 7,9.2 Pharmacodynamic Analysis

Not applicable.

#### 7.10 Other Outcomes

Not applicable.

#### **Safety Analysis** 7.11

#### 7.11.1 Adverse Events

7.11.1.1 Overview of Treatment-Emergent Adverse Events

Analysis Set:

Analysis

Variable(s):

Analytical


Method(s):

- The following summaries will be provided.

  (1) Overview of Treatment-Emergent Adverse Events

  1) Any adverse event

  2) Grade 3 or higher adverse event

  3) Drug-related adverse event

  4) Drug-related grade 3 or 1

  5) Serious advers

  6) Drug-

  - 6) Drug-related serious adverse event
  - 7) Adverse events resulting in any study drug dose reduction
  - 8) Adverse events resulting in any study drug dose modification
  - 9) Adverse events resulting in any study drug discontinuation
  - 10) On-study deaths

For summary 8), dose modification will include dose reduction, dose increase, dose delay, and dose discontinuation.

TEAEs will be counted according to the rules below.

#### Number of subjects

Summaries for 3), 4), and 6)

A subject with occurrences of TEAE in both categories (i.e., Related and Not Related) will be counted once in the Related category.

Summaries for 2) and 4)

A subject with multiple occurrences of TEAE will be counted once for the TEAE with the maximum intensity.

• Summaries other than 2), 3), 4), and 6) A subject with multiple occurrences of TEAE will be counted only once.

## 7.11.1.2 Overview of Treatment-Emergent Adverse Events by Subgroups

Safety Analysis Set Analysis Set:

Analysis

Variable(s): **TEAE** 

[1-6, 7-12, 13-18, >=19]Subgroup(s): Cycles

> Sex [Male, Female]

[Min<= - <30, 30<= - <60, Creatinine Clearance (mL/min)

Analytical

The same overview summary as Section 7.11.1.1 will be provided for each Method(s): subgroup category.

- (1) Overview of Treatment-Emergent Adverse Events by Cycle in Subjects with >= 12 Cycles Exposure
- (2) Overview of Treatment-Emergent Adverse Events by Sex
- (3) Overview of Treatment-Emergent Adverse Events by Creatinine Clearance

The summary in (1) will be based on subjects who have completed 12 cycles or more of the study drug

## 7.11.1.3 Displays of Treatment-Emergent Adverse events

Analysis Set: Safety Analysis Set

Analysis

Variable(s):

Categories: Intensity [Grade 1, Grade 2, Grade 3, Grade 4,

Grade 5]

Time of Onset (Cycle) [1-3, 4-6, 7-9, 10-12, 13-15,

16 - 18, 19 - 21, 22 - 24

Analytical
Method(s): The following summaries will be provided using frequency distribution.

TEAEs will be coded using the MedDRA and will be summarized using

SOC, HLT, and PT.

SOC, HLT, and PT will be sorted in decreasing frequency for tables provided by SOC, HLT, and PT. SOC will be sorted alphabetically and PT will be sorted in decreasing frequency for tables provided by SOC and PT. PT will be sorted in decreasing frequency for tables provided by PT only.

Property of Takeda.

- (1) Treatment-Emergent Adverse Events by System Organ Class, High Level Term, and Preferred Term
- (2) Treatment-Emergent Adverse Events by Preferred Term
- cerms of Use (3) Treatment-Emergent Drug-Related Adverse Events by System Organ Class, High Level Term, and Preferred Term
- (4) Treatment-Emergent Grade 3 or Higher Adverse Events by System Organ Class, High Level Term, and Preferred Term
- (5) Treatment-Emergent Grade 3 or Higher Adverse Events by Preferred Term
- (6) Treatment-Emergent Drug-Related Grade 3 or Higher Adverse Events by System Organ Class, High Level Term, and Preferred Term
- (7) Treatment-Emergent Grade 4 Adverse Events by System Organ Class, High Level Term, and Preferred Term
- (8) Intensity of Treatment-Emergent Adverse Events by System Organ Class, High Level Term, and Preferred Term
- (9) Intensity of Treatment-Emergent Drug-Related Adverse Events by System Organ Class, High Level Term, and Preferred Term
- (10) Treatment-Emergent Adverse Events Leading to Study Drug Discontinuation by System Organ Class, High Level Term, and Preferred Term
- (11) Treatment-Emergent Serious Adverse Events by System Organ Class, High Level Term, and Preferred Term
- (12) Treatment-Emergent Drug-Related Serious Adverse Events by System Organ Class, High Level Term, and Preferred Term
- (13) Treatment-Emergent Adverse Events by System Organ Class, High Level Term, and Preferred Term Over Time
- (14) Most Frequent Non Serious Treatment-Emergent Adverse Events by System Organ Class and Preferred Term
- (15) Summary of Treatment-Emergent Adverse Events which Resulted in Dose Reduction by System Organ Class and Preferred Term
- (16) Summary of Treatment-Emergent Adverse Events which Resulted in Dose Held by System Organ Class and Preferred Term
- (17) Summary of Treatment-Emergent Adverse Events which Resulted in Dose Discontinuation by System Organ Class and Preferred Term The frequency distribution will be provided according to the rules below. Number of subjects

ns of Use

- Summary tables other than (4) to (9) and (13)

  A subject with multiple occurrences of TEAE within a SOC will be counted only once in that SOC. A subject with multiple occurrences of TEAE within an HLT will be counted only once in that HLT. A subject with multiple occurrences of TEAE within a PT will be counted only once in that PT. Percentages will be based on the number of subjects in the safety analysis set.
- Summary tables for (4) to (9)
  A subject with multiple occurrences of TEAE within a SOC, an HLT, or a
  PT will be counted only once for the TEAE with the maximum intensity.
  Percentages will be based on the number of subjects in the safety analysis set.
- Summary table for (13)

A subject with a TEAE that occurs in more than one interval is counted in all the intervals that the TEAE occurs. For each time interval, a subject with multiple occurrences of TEAE within a SOC, an HLT, or a PT will be counted only once in that SOC, HLT, or PT.

When calculating percentages for each time interval, the number of subjects at risk (i.e., subjects who either have an exposure or have an occurrence of TEAE, during or after the corresponding time interval) will be used as the denominator. The number of subjects whose onset of any one of the TEAEs is within the time interval will be used as the numerator.

- Summary table for (14)
   Most frequent non-serious TEAEs refer to PTs that are not serious whose percentages are at least 5%.
- Summary table for (15)
  TEAEs which resulted in dose reduction in Ixazomib, in Lenalidomide, and in Dexamethasone will each be displayed, as well as the TEAEs which resulted in dose reduction in any of Ixazomib, Lenalidomide, or Dexamethasone.
- Summary table for (16)
   TEAEs which resulted in dose held in Ixazomib, in Lenalidomide, and in Dexamethasone will each be displayed, as well as the TEAEs which resulted in dose held in any of Ixazomib, Lenalidomide, or Dexamethasone.
- Summary table for (17)

Probeity of Lakeda.

Analysis Set: Safety Analysis Set
Analysis
Variable(s): TEAE of clinical importance
Treatment-emergent haemorrhage adverse events

NCI CTCAE Grade

[Grade 1 G- '
Indicate the displayed, as well as

Lenatidomide, or Dexamethasone.

7.11.1.4 Displays of Treatment-Emergent Adverse Events of Clinical Importance and Haemorrhage

Analysis Set: Safety Analysis Set

Analysis

Variable(s): TEAE of clinical importance

Treatment-emergent haemorrhage adverse events

Categories: NCI CTCAE Grade

[Grade 1 G- '
Inalytical

[fethod(s): A' '

Adverse events of clinical importance will include diarrhea, rash, Method(s):

neutropenia, thrombocytopenia, nausea, peripheral neuropathy, vomiting, arrhythmias, renal, liver impairment, hypotension, heart failure, new primary malignancy, myocardial infarction, and encephalopathy. The following summaries will be provided using frequency distribution. For (2) and (3), descriptive statistics will be provided. For (3), time to resolution from the first onset of the AE will be summarized. If no date of resolution is recorded, then the last date of visit will be used as the date of resolution.

TEAEs will be coded using the MedDRA and will be summarized using PT for (1) to (6). For (1), PT will be sorted in decreasing frequency. For (4) to (6), AECI and PT will both be sorted alphabetically. A subject with multiple occurrences of TEAE within a PT will be counted only once for the TEAE with the maximum intensity. For (4), TEAEs of clinical importance which resulted in dose reduction in Ixazomib, in Lenalidomide, and in Dexamethasone will each be displayed, as well as TEAEs of clinical importance which resulted in dose reduction in any of Ixazomib, Lenalidomide, or Dexamethasone. For (5), TEAEs of clinical importance which resulted in dose held in Ixazomib, in Lenalidomide, and in Dexamethasone will each be displayed, as well as TEAEs of clinical importance which resulted in dose held in any of Ixazomib, Lenalidomide, or Dexamethasone. For (6), TEAEs of clinical importance which resulted in

dose discontinuation in Ixazomib, in Lenalidomide, and in Dexamethasone

750 (15E

will each be displayed, as well as TEAEs of clinical importance which resulted in dose discontinuation in any of Ixazomib, Lenalidomide, or Dexamethasone. For (7), TEAEs will be summarized using SOC, HLT, and PT, where SOC, HLT, and PT will be sorted in decreasing frequency. TEAEs will be graded using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) (Version 4.03).

- (1) Treatment-Emergent Adverse Events of Clinical Importance by Preferred Term and NCI CTCAE Grade
- (2) Summary of Time to First Onset in Treatment-Emergent Adverse Events of Clinical Importance
- (3) Summary of Time to Resolution in Treatment-Emergent Adverse Events of Clinical Importance
- (4) Treatment-Emergent Adverse Events of Clinical Importance which Resulted in Dose Reduction by Preferred Term
- (5) Treatment-Emergent Adverse Events of Clinical Importance which Resulted in Dose Held by Preferred Term
- (6) Treatment-Emergent Adverse Events of Clinical Importance which Resulted in Dose Discontinuation by Preferred Term
- (7) Treatment-Emergent Haemorrhage Adverse Events by System Organ Class, High Level Term, and Preferred Term

7.11.1.5 Summary of Treatment-Emergent Adverse Events Overall, and by Toxicity, Seriousness, Relatedness, Discontinuation, and Dose Modification

Analysis Set: Safety Analysis Set

Analysis

Variable(s): TEAE

TEAE of clinical importance

Analytical

Method(s):

The following summaries will be provided using frequency distribution. The summaries will include the number and percentages of subjects who had any TEAEs, drug-related TEAEs, Grade 3 or higher TEAEs, Grade 3 or higher drug-related TEAEs, serious TEAEs, TEAEs resulting in death, TEAEs leading to study drug discontinuation, TEAEs which resulted in dose reduction, dose held, and dose delayed in any of Ixazomib, Lenalidomide, or Dexamethasone. TEAEs will be coded using the MedDRA and will be

summarized using SOC and PT. SOC and PT will be sorted in decreasing frequency.

- (1) Summary of Treatment-Emergent Adverse Events Overall, and by Toxicity, Seriousness, Relatedness, Discontinuation, and Dose Modification
- (eins of Use (2) Summary of Treatment-Emergent Adverse Events of Clinical Importance ating applifect to the applif Overall, and by Toxicity, Seriousness, Relatedness, Discontinuation, and Dose Modification

#### 7.11.2 Clinical Laboratory Evaluations

#### 7.11.2.1 Hematology and Blood Chemistry

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Hematology

> Hematocrit Platelet Count Hemoglobin Neutrophils **WBC** Count Lymphocytes

Serum Chemistry

Blood Urea Nitrogen Creatinine Total Bilirubin

Uric Acid Alkaline Phosphatase Lactate dehydrogenase

(LDH)

**AST ALT** Albumin Potassium Glucose Sodium Chloride Carbon dioxide Magnesium

Calcium Phosphate Thyroid Stimulating

Hormone (TSH)

Categories: Intensity [Grade 0, Grade 1, Grade 2, Grade 3, Grade 4]

Hematology: Screening, Baseline, Cycle 1 Day 1, Cycle 1 Day 7, Cycle 1

Day 14, Cycle 1 Day 21, Cycle 2 Day 1, Cycle 2 Day 7, Cycle 2 Day 14,

Cycle 2 Day 21, Cycle 3 Day 1, Cycle 3 Day 14, Cycle 4 Day 1, Cycle 5 Day

1, Cycle 6 Day 1, ... (up to the maximum cycle), End of Treatment, Last

Assessment

Serum Chemistry: Screening, Baseline, Cycle 1 Day 1, Cycle 2 Day 1, Cycle

3 Day 1, Cycle 4 Day 1, Cycle 5 Day 1, Cycle 6 Day 1, ... (up to the

maximum cycle), End of Treatment, Last Assessment

Analytical

Method(s): For each variable, (1) will be provided.

For applicable variables, (2), (3), and (4) will be provided.

NCI CTCAE (Version 4.03) will be used for grading. Last Assessment is defined as the last measurement prior to or on the last visit conducted 30 days after the last dose of study drug regimen.

Laboratory test results from the central laboratory will be used when they are available. Laboratory test results from local laboratory will be used only when no central laboratory test result exists at the same scheduled sample collection time point.

- (1) Summary of Laboratory Test Results and Change from Baseline by Visit Descriptive statistics for observed values for each visit and changes from baseline will be provided.
- (2) Case Plots
  Plots over time for each subject will be presented for platelet count and neutrophils.
- (3) Line Plot of Platelet Count Over Time

  For the platelet count, the overall median over time will be presented.
- (4) Maximum Grade Shift from Baseline of Laboratory Parameters

  The maximum (worst) post-baseline grade will be determined for each subject. Shift tables showing the number of subjects in each grade category at baseline and post-baseline visit will be provided using evaluable data.

## 7.11.3 Vital Signs and Weight

Analysis Set: Safety Analysis Set

Analysis

Variable(s): Systolic Blood Pressure (mmHg)

Diastolic Blood Pressure (mmHg)

Heart Rate (bpm)

Respiratory Rate (bpm)

Temperature (C)

Weight (kg)

Visit: Screening, Baseline, Cycle 1 Day 1, Cycle 2 Day 1, Cycle 3 Day 1,

Cycle 4 Day 1, ... (up to the maximum cycle), End of Treatment,

Last Assessment

#### Analytical

Method(s):

as the last measurement prior to or on the last conducted 30 days after the last dose of study drug regimen.

(1) Summary of Vital Signs Parameters and Change from Baseline by Visit Descriptive statistics for observed values for each visit and change baseline will be provided. and subject to the applicable

#### 7.11.4 12-Lead ECGs

Not applicable.

#### 7.11.5 Other Observations Related to Safety

#### 7.11.5.1 ECOG Performance Status

Safety Analysis Set Analysis Set:

Analysis

**ECOG Performance Status** Variable(s):

Categories: **ECOG Score** 

Screening, Baseline, Cycle 2 Day 1, Cycle 3 Day 1, ... (up to the maximum Visit:

cycle), End of Treatment, Last Assessment

Analytical

For each variable, the following summaries will be provided. Method(s):

> Last Assessment is defined as the last measurement prior to or on the last visit conducted 30 days after the last dose of study drug regimen.

(1) ECOG Performance Status Data Measured Over Time

Descriptive statistics for observed values for each visit and changes from baseline will be provided.

(2) ECOG Performance Score Shift from Baseline to Post-Baseline Assessments Over Time

Shift tables showing the number of subjects in each ECOG score category at baseline and each post-baseline visit will be provided.

#### 7.11.5.2 Subsequent Anti-Cancer Therapy

Safety Analysis Set

Analysis

Variable(s): Subsequent Anti-Cancer Therapy

Analytical

DIE Terms of Use Method(s): (1) Subsequent Anti-Cancer Therapy by Class of Agent and WHO Generic Term

Frequency distributions will be provided.

#### 7.12 **Interim Analysis**

Analysis is planned to be performed twice during the study. The primary analysis is planned to be performed using the data obtained at approximately 12 months from the enrollment of the last patient. The final analysis is planned to be performed after the final database lock using the data obtained at approximately 24 months from the enrollment of the last patient. The timing of analysis may be changed or additional analysis may be added upon request of the regulatory authorities.

#### **Changes in the Statistical Analysis Plan** 7.13

Property of Takeda. For non-commercial use only all The analyses in the statistical analysis plan do not differ from the analyses specified in the